CLINICAL TRIAL: NCT00420238
Title: A Multicentre, Double-Blind, Placebo-Controlled, Randomised Study of Etanercept in the Treatment of Adult Patients With Active, Severe, and Advanced Axial Ankylosing Spondylitis
Brief Title: Study Evaluating Etanercept for the Treatment of Active, Severe, and Advanced Axial Ankylosing Spondylitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0881A3-403
Record Dates: First submitted 2007-01-08; First posted 2007-01-11 (Estimated); Results first posted 2010-06-15 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Ankylosing Spondylitis
Keywords: Axial Ankylosing Spondylitis; Adult
MeSH Terms: conditions — Spondylitis, Ankylosing | interventions — Etanercept

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Experimental)
  Interventions: Drug: Etanercept (Enbrel)
- B (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Etanercept (Enbrel) — 50 mg injection once weekly
  Arms: A
Other: Placebo — placebo
  Arms: B

SUMMARY:
Evaluation of the efficacy and safety of etanercept (Enbrel) in patients with active, severe and advanced ankylosing spondylitis.

ELIGIBILITY:
Inclusion criteria

* Active and severe ankylosing spondylitis
* Ankylosing spondylitis refractory to standard anti-rheumatic treatment
* Between 18 and 70 years of age

Exclusion criteria

* Prior exposure to any TNF-inhibitor, including etanercept
* DMARDs (other than hydroxychloroquine, methotrexate and sulphasalazine) within 4 weeks of study drug initiation
* Dose of NSAIDs changed within two weeks of study drug initiation

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2007-01; Primary Completion 2009-02 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer; Trial Manager, Principal Investigator — For France, infomedfrance@wyeth.com; Trial Manager, Principal Investigator — For Germany, medinfoDEU@wyeth.com; Trial Manager, Principal Investigator — For Netherlands, trials-NL@wyeth.com; Trial Manager, Principal Investigator — For Hungary: WPBUMED@wyeth.com
Locations (21):
- France (16):
  - Amiens
  - Arles
  - Avignon
  - Bordeaux
  - Cabestany
  - Corbeil-Essonnes
  - Montpellier
  - Nice
  - Orléans
  - Paris (Ambroise Pare)
  - Paris (Bichat)
  - Paris (cochin)
  - Paris (Pitie Salpetriere)
  - Paris (Saint Antoine)
  - Strasbourg
  - Toulouse
- Germany (2):
  - Berlin
  - Herne
- Hungary (2):
  - Budapest
  - Debrecen
- Maastricht, Netherlands

REFERENCES:
- [Derived] Dougados M, Braun J, Szanto S, Combe B, Geher P, Leblanc V, Logeart I. Continuous efficacy of etanercept in severe and advanced ankylosing spondylitis: results from a 12-week open-label extension of the SPINE study. Rheumatology (Oxford). 2012 Sep;51(9):1687-96. doi: 10.1093/rheumatology/kes125. Epub 2012 May 30. PMID 22653382
- [Derived] Dougados M, Braun J, Szanto S, Combe B, Geher P, Leblanc V, Logeart I. Nonsteroidal antiinflammatory drug intake according to the Assessment of SpondyloArthritis International Society Score in clinical trials evaluating tumor necrosis factor blockers: example of etanercept in advanced ankylosing spondylitis. Arthritis Care Res (Hoboken). 2012 Feb;64(2):290-4. doi: 10.1002/acr.20671. PMID 22006544
- [Derived] Dougados M, Braun J, Szanto S, Combe B, Elbaz M, Geher P, Thabut G, Leblanc V, Logeart I. Efficacy of etanercept on rheumatic signs and pulmonary function tests in advanced ankylosing spondylitis: results of a randomised double-blind placebo-controlled study (SPINE). Ann Rheum Dis. 2011 May;70(5):799-804. doi: 10.1136/ard.2010.139261. Epub 2011 Feb 13. PMID 21317434

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects with advanced ankylosing spondylitis (AS) by Modified New York criteria, advanced and severe disease with intervertebral bridges, and an axial defined by a score of ≥30 for overall level of AS neck, back, or hip pain on the BASDAI were eligible to participate in the study and were randomized at 19 study sites.
Pre-assignment Details: Subjects completed a screening period of up to 6 weeks duration prior to entering the treatment period; 95 subjects were screened, and 82 subjects were randomized.
Groups:
- Etanercept/Etanercept: Etanercept 50 mg subcutaneously (SC) once weekly
- Placebo/Etanercept: Placebo subcutaneously (SC), once weekly; Etanercept 50 mg SC, once weekly
Period: 12 Week Double-Blind Treatment Period 1
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Started | 39 | 43
Completed | 38 | 39
Not Completed | 1 | 4
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal of Consent | 0 | 1
Period: 12 Week Open-Label Treatment Period 2
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Started | 38 | 39
Completed | 36 | 38
Not Completed | 2 | 1
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal of Consent | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Etanercept: 50 mg subcutaneously (SC), once weekly
- Placebo: Subcutaneously (SC), once weekly
- Total: Total of all reporting groups
Arm/Group | Etanercept | Placebo | Total
Number analyzed (Participants) | 39 | 43 | 82
Age Continuous [Mean (Standard Deviation); unit: years] | 46.2 (10.8) | 48.2 (47.3) | 47.3 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 37 | 39 | 76

OUTCOME MEASURES:

1. Primary Outcome: Normalized Net Incremental Area Under the Curve (AUC) for the Bath Ankylosing Spondylitis Disease Activities Index (BASDAI) Between Randomization and Week 12
Description: BASDAI subject asessment of discomfort, pain and fatigue measured using a 100 millimeter Visual Analog Scale; range: 0=none to 100=very severe. Normalized net incremental area under the curve (AUC) = area between baseline and the BASDAI curve as a function of time (randomization to Week 12); computed using the linear trapezoidal method. All areas above baseline and under the curve are positive and all areas below baseline and above the curve are negative. Net incremental AUC = sum of these areas; this result was then divided by the study duration of the patients; negative value = improvement.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: Modified Intent-To-Treat (mITT) population: includes all randomized subjects who received at least 1 dose of blinded study drug. Last observation carried forward (LOCF).
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
millimeters | -19.79 (16.83) [-25.03 to -14.54] | -10.96 (16.46) [-15.95 to -5.97]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Comparison of least squares means. Primary analysis: analysis of covariance (ANCOVA) with treatment as a factor and BASDAI baseline as a covariate; Test type: Superiority or Other; p = 0.019, ANCOVA; Mean Difference (Final Values) = -8.83, 95% CI 2-sided [-16.5 to -1.51] — Least squares mean difference = mean difference final value

2. Secondary Outcome: Percent of Subjects Achieving Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) 50 Response
Description: BASDAI subject assessment of discomfort, pain and fatigue was measured using a 100 millimeter Visual Analog Scale (VAS); range: 0=none to 100=very severe. BASDAI 50 response defined as at least a 50 percent (%) improvement (decrease) from baseline to observation (last observation carried forward) in the BASDAI. Baseline score minus score at observation divided by Baseline score * 100 = >=50%.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF.
Measure: Number; unit: percent of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
percent of participants
  Week 2 | 23.08 | 9.30
  Week 4 | 28.21 | 16.28
  Week 8 | 41.03 | 23.26
  Week 12 | 46.15 | 23.26
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Week 2: Generalized estimating equations (GEE) model, using a logit link, a binomial distribution and an auto-regressive correlation structure, with treatment groups, visits and their interactions as fixed factors; Test type: Superiority or Other; p = 0.098, GEE model; Odds Ratio (OR) = 2.92, 95% CI 2-sided [0.82 to 10.42] — An odds-ratio greater than 1 indicates the odds of response is greater in the etanercept group than in the placebo group
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Week 4: Generalized estimating equations (GEE) model, using a logit link, a binomial distribution and an auto-regressive correlation structure, with treatment groups, visits and their interactions as fixed factors; Test type: Superiority or Other; p = 0.197, GEE model; Odds Ratio (OR) = 2.02, 95% CI 2-sided [0.69 to 5.88] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; Week 8: Generalized estimating equations (GEE) model, using a logit link, a binomial distribution and an auto-regressive correlation structure, with treatment groups, visits and their interactions as fixed factors; Test type: Superiority or Other; p = 0.087, GEE model; Odds Ratio (OR) = 2.30, 95% CI 2-sided [0.89 to 5.95] — [estimate comment as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; Week 12: Generalized estimating equations (GEE) model, using a logit link, a binomial distribution and an auto-regressive correlation structure, with treatment groups, visits and their interactions as fixed factors; Test type: Superiority or Other; p = 0.031, GEE model; Odds Ratio (OR) = 2.83, 95% CI 2-sided [1.10 to 7.29] — [estimate comment as in outcome 2, analysis 1]

3. Secondary Outcome: Percent of Subjects Achieving Assessment Ankylosing Spondylitis (ASAS) 20 at Weeks 2, 4, 8, 12
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) patients; 4 domains: patient global assessment of disease activity, pain, function,and inflammation. ASAS 20 = 20% improvement (versus baseline) and an absolute change (net improvement) ≥ 10 millimeters (mm) on a 0-100 mm scale (100=high disease activity) for ≥ 3 domains, and no worsening (absence of deterioration by >=20% and by >= 10 mm) in remaining domain.
Time Frame: Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF.
Measure: Number; unit: percent of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
percent of participants
  Week 2 | 30.77 | 20.93
  Week 4 | 41.03 | 30.23
  Week 8 | 64.10 | 27.91
  Week 12 | 66.67 | 32.56
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Week 2: Generalized estimating equations (GEE) model, using a logit link, a binomial distribution and an auto-regressive correlation structure, with treatment groups, visits, and their interaction as fixed factors; Test type: Superiority or Other; p = 0.310, GEE model; Odds Ratio (OR) = 1.68, 95% CI 2-sided [0.62 to 4.57] — An odds ratio greater than 1 indicates the odds of response is greater in the etanercept group than in the placebo group
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Week 4: Generalized estimating equations (GEE) model, using a logit link, a binomial distribution and an auto-regressive correlation structure, with treatment groups, visits, and their interaction as fixed factors; Test type: Superiority or Other; p = 0.309, GEE model; Odds Ratio (OR) = 1.61, 95% CI 2-sided [0.65 to 3.99] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: Etanercept vs Placebo; Week 8: Generalized estimating equations (GEE) model, using a logit link, a binomial distribution and an auto-regressive correlation structure, with treatment groups, visits, and their interaction as fixed factors; Test type: Superiority or Other; p = 0.001, GEE model; Odds Ratio (OR) = 4.61, 95% CI 2-sided [1.81 to 11.74] — [estimate comment as in outcome 3, analysis 1]
Statistical Analysis 4: Comparison: Etanercept vs Placebo; Week 12: Generalized estimating equations (GEE) model, using a logit link, a binomial distribution and an auto-regressive correlation structure, with treatment groups, visits, and their interaction as fixed factors; Test type: Superiority or Other; p = 0.003, GEE model; Odds Ratio (OR) = 4.14, 95% CI [1.65 to 10.42] — [estimate comment as in outcome 3, analysis 1]

4. Secondary Outcome: Percent of Subjects Acheiving Assessment Ankylosing Spondylitis (ASAS) 20 at Weeks 14, 18, 24
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) patients; 4 domains: patient global assessment of disease activity, pain, function, and inflammation. ASAS 20 = 20% improvement (versus baseline) and an absolute change (net improvement) ≥ 10 units (millimeters) on a 0-100 scale (100=high disease activity) for ≥ 3 domains, and no worsening (absence of deterioration by >=20% and by >=10 mm) in remaining domain.
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population: all subjects who received at least 1 dose of open test article (Etanercept). LOCF.
Measure: Number; unit: percent of participants
Groups:
- Etanercept/Etanercept: Double-blind Period 1: Etanercept 50 mg subcutaneously (SC) once weekly; Open-label Period 2: etanercept 50 mg subcutaneously (SC), once weekly
- Placebo/Etanercept: Double-blind Period 1: placebo subcutaneously (SC), once weekly; Open-label Period 2: etanercept subcutaneously (SC), once weekly
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
percent of participants
  Week 14 | 71.05 | 53.85
  Week 18 | 71.05 | 64.10
  Week 24 | 84.21 | 66.67

5. Secondary Outcome: Percent of Subjects Achieving Assessment Ankylosing Spondylitis (ASAS) 50 at Weeks 2, 4, 8, 12
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) patients; 4 domains: patient global assessment of disease activity, pain, function, inflammation. ASAS 50 = 50% improvement (versus baseline) and an absolute (net) change ≥ 20 units on a 0-100 scale (high disease activity) for ≥ 3 domains, and no worsening (absence of deterioration by >=20% and by >=10 mm) in remaining domain.
Time Frame: Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF.
Measure: Number; unit: percent of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
percent of participants
  Week 2 | 17.95 | 9.30
  Week 4 | 23.08 | 16.28
  Week 8 | 35.90 | 16.28
  Week 12 | 38.46 | 13.95
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.259, GEE model; Odds Ratio (OR) = 2.13, 95% CI 2-sided [0.57 to 7.94] — An odds ratio greater than 1 indicates the odds of response is greater in etanercept group than in placebo group
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.440, GEE model; Odds Ratio (OR) = 1.54, 95% CI [0.51 to 4.64] — An odds ratio greater than 1 indicates the odds of response is greater in etanercept group than in placebo group
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.046, GEE model; Odds Ratio (OR) = 2.88, 95% CI [1.02 to 8.16] — An odds ratio greater than 1 indicates the odds of response is greater in etanercept group than in placebo group
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.014, GEE model; Odds Ratio (OR) = 3.85, 95% CI [1.31 to 11.32] — An odds ratio greater than 1 indicates the odds of response is greater in etanercept group than in placebo group

6. Secondary Outcome: Percent of Subjects Achieving Assessment Ankylosing Spondylitis (ASAS) 50 at Weeks 14, 18, 24
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) patients; 4 domains: patient global assessment of disease activity, pain, function, inflammation. ASAS 50 = 50% improvement (vs. baseline) and an absolute (net) change ≥ 20 units on a 0-100 scale (high disease activity) for ≥ 3 domains, and no worsening (absence of deterioration by >=20% and by >=10 mm) in remaining domain.
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; LOCF.
Measure: Number; unit: percent of particpants
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
percent of particpants
  Week 14 | 44.74 | 43.59
  Week 18 | 50.00 | 48.72
  Week 24 | 60.53 | 51.28

7. Secondary Outcome: Percent of Subjects Achieving Assessment Ankylosing Spondylitis (ASAS) 70 at Weeks 2, 4, 8, 12
Description: ASAS measures symptomatic improvement in Ankylosing Spondylitis (AS) patients; 4 domains: patient global assessment of disease activity, pain, function, inflammation. ASAS 70 = 70% improvement (vs. baseline) and an absolute change ≥ 20 units on a 0-100 scale (high disease activity) for ≥ 3 domains, and no worsening (absence of deterioration by >=20% and by >= 10 mm) in remaining domain.
Time Frame: Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF.
Measure: Number; unit: percent of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
percent of participants
  Week 2 | 12.82 | 4.65
  Week 4 | 17.95 | 4.65
  Week 8 | 15.38 | 4.65
  Week 12 | 25.64 | 9.30
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.204, GEE model; Odds Ratio (OR) = 3.01, 95% CI 2-sided [0.55 to 16.53] — An odds ratio greater than 1 indicates the odds of response is greater in etanercept group than in placebo group
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.073, GEE model; Odds Ratio (OR) = 4.48, 95% CI [0.87 to 23.07] — An odds ratio greater than 1 indicates the odds of response is greater in etanercept group than in placebo group
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.121, GEE model; Odds Ratio (OR) = 3.73, 95% CI [0.71 to 19.69] — An odds ratio greater than 1 indicates the odds of response is greater in etanercept group than in placebo group
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.058, GEE model; Odds Ratio (OR) = 3.36, 95% CI [0.96 to 11.80] — An odds ratio greater than 1 indicates the odds of response is greater in etanercept group than in placebo group

8. Secondary Outcome: Percent of Subjects Achieiving Assessment Ankylosing Spondylitis (ASAS) 70 at Weeks 14, 18, 24
Description: as for outcome 7
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; LOCF.
Measure: Number; unit: percent of participants
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
percent of participants
  Week 14 | 31.58 | 33.33
  Week 18 | 31.58 | 30.77
  Week 24 | 36.84 | 35.90

9. Secondary Outcome: Percent of Subjects Achieving Partial Remission at Weeks 2, 4, 8, 12
Description: Partial remission defined as a score of <20 millimeters (mm) on a scale of 0 to 100 mm in each of 4 domains: Visual Analog Scale (VAS) patient global assessment, VAS pain score (Total Back Pain), Bath Ankylosing Spondylitis Functional Index (BASFI) score, and Bath Ankylosing Spondylitis Disease Activities Index (BASDAI)-mean of two morning stiffness-related VAS scores. A negative score indicates an improvement in disease activity and a positive score indicates worsening.
Time Frame: Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF.
Measure: Number; unit: percent of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
percent of participants
  Week 2 | 7.69 | 2.33
  Week 4 | 10.26 | 2.33
  Week 8 | 17.95 | 4.65
  Week 12 | 17.95 | 4.65
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.287, GEE model; Odds Ratio (OR) = 3.50, 95% CI 2-sided [0.35 to 35.14] — An odds ratio greater than 1 indicates the odds of response is greater in etanercept group than in placebo group
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 3, analysis 2]; Test type: Superiority or Other; p = 0.169, GEE model; Odds Ratio (OR) = 4.80, 95% CI [0.51 to 44.94] — An odds ratio greater than 1 indicates the odds of response is greater in etanercept group than in placebo group
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 3, analysis 3]; Test type: Superiority or Other; p = 0.073, GEE model; Odds Ratio (OR) = 4.48, 95% CI [0.87 to 23.07] — An odds ratio greater than 1 indicates the odds of response is greater in etanercept group than in placebo group
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 3, analysis 4]; Test type: Superiority or Other; p = 0.073, GEE model; Odds Ratio (OR) = 4.48, 95% CI [0.87 to 23.07] — An odds ratio greater than 1 indicates the odds of response is greater in etanercept group than in placebo group

10. Secondary Outcome: Percent of Subjects Achieving Partial Remission at Weeks 14, 18, 24
Description: as for outcome 9
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; LOCF.
Measure: Number; unit: percent of participants
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
percent of participants
  Week 14 | 28.95 | 23.08
  Week 18 | 31.58 | 25.64
  Week 24 | 28.95 | 23.08

11. Secondary Outcome: Normalized Net Incremental Area Under the Curve (AUC) for Patient Global Assessment (PGA) Between Baseline and Week 12
Description: PGA was measured using a 100 millimeter Visual Analog Scale (VAS) ranging from 0 = very good to 100 = very bad. Normalized net incremental area under the curve (AUC)=area between baseline and the Patient Global Asessment curve as a function of time (randomization to Week 12); computed using the linear trapezoidal method. All areas above baseline and under the curve are positive and all area below baseline and above the curve are negative. Net incremental AUC = sum of these areas; this result was then divided by the study duration of the patients; negative value = improvement.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF. N = number of subjects with evaluable data.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 41
millimeters | -20.35 [-26.23 to -14.47] | -10.39 [-16.13 to -4.66]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Analysis of covariance (ANCOVA) with treatment as a factor and baseline value as a covariate; Test type: Superiority or Other; p = 0.018, ANCOVA; Mean Difference (Final Values) = -9.95, 95% CI 2-sided [-18.19 to -1.72] — Least squares mean difference = mean difference final value

12. Secondary Outcome: Change From Baseline in Patient Global Assessment Visual Analog Scale (VAS) at Weeks 2, 4, 8, 12
Description: Patient global assessment of all the ways ankylosing spondylitis affected them in the last 48 hours using a 100 millimeter (mm) Visual Analog Scale (VAS); range 0=very good to 100=very bad.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
units on scale
  Week 2 | -16.90 [-23.96 to -9.85] | -8.36 [-15.24 to -1.49]
  Week 4 | -19.06 [-26.11 to -12.01] | -11.04 [-17.92 to -4.16]
  Week 8 | -25.29 [-32.35 to -18.24] | -10.56 [-17.44 to -3.68]
  Week 12 | -25.79 [-32.84 to -18.74] | -16.52 [-23.40 to -9.64]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Week 2: Comparison of leasts squares means. Mixed-model analysis of covariance (ANCOVA) using an auto-regressive correlation structure with treatment groups, visits and their interaction as fixed factors, baseline value as a covariate, and patients as a random factor; Test type: Superiority or Other; p = 0.089, ANCOVA; Mean Difference (Final Values) = -8.54, 95% CI 2-sided [-18.40 to 1.33] — Least squares mean difference = mean difference final value
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Week 4: Comparison of leasts squares means. Mixed-model analysis of covariance (ANCOVA) using an auto-regressive correlation structure with treatment groups, visits and their interactions as fixed factors, baseline value as a covariate, and patients as a random factor; Test type: Superiority or Other; p = 0.110, ANCOVA; Mean Difference (Final Values) = -8.02, 95% CI [-17.89 to 1.85] — Least squares mean difference = mean difference final value
Statistical Analysis 3: Comparison: Etanercept vs Placebo; Week 8: Comparison of leasts squares means. Mixed-model analysis of covariance (ANCOVA) using an auto-regressive correlation structure with treatment groups, visits and their interactions as fixed factors, baseline value as a covariate, and patients as a random factor; Test type: Superiority or Other; p = 0.004, ANCOVA; Mean Difference (Final Values) = -14.73, 95% CI [-24.60 to -4.86] — Least squares mean difference = mean difference final value
Statistical Analysis 4: Comparison: Etanercept vs Placebo; Week 12: Comparison of leasts squares means. Mixed-model analysis of covariance (ANCOVA) using an auto-regressive correlation structure with treatment groups, visits and their interactions as fixed factors, baseline value as a covariate, and patients as a random factor; Test type: Superiority or Other; p = 0.065, ANCOVA; Mean Difference (Final Values) = -9.27, 95% CI [-19.14 to 0.59] — Least squares mean difference = mean difference final value

13. Secondary Outcome: Change From Baseline in Patient Global Assessment at Weeks 14, 18, 24
Description: as for outcome 12
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; LOCF.
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
units on scale
  Week 14 | -31.26 [-40.35 to -22.18] | -31.20 [-40.57 to -21.83]
  Week 18 | -35.50 [-44.18 to -26.82] | -31.92 [-41.44 to -22.40]
  Week 24 | -40.70 [-49.18 to -32.23] | -34.19 [-42.86 to -25.53]

14. Secondary Outcome: Normalized Net Incremental Area Under the Curve (AUC) for Physician Global Assessment (PGA) Between Baseline and Week 12
Description: PGA was measured using a 100 millimeter Visual Analog Scale (VAS) ranging from 0 = very good to 100 = very bad. Normalized net incremental area under the curve (AUC) = area between baseline and the Physician Global Assessment curve as a function of time (randomization to Week 12); computed using the linear trapezoidal method. All areas above baseline and under the curve are positive and all area below baseline and above the curve are negative. Net incremental AUC = sum of these areas; this result was then divided by the study duration of the patients; negative value = improvement.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF. N= number of subjects with evaluable data.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 42
millimeters | -24.14 [-28.97 to -19.32] | -13.15 [-17.80 to -8.50]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Analysis of covariance (ANCOVA) with treatment as a factor and baseline value as a covariate; Test type: Superiority or Other; p = 0.002, ANCOVA; Mean Difference (Final Values) = -10.99, 95% CI 2-sided [-17.70 to -4.28] — Least squares mean difference = mean difference final value

15. Secondary Outcome: Change From Baseline in Physician Global Assessment Visual Analog Scale at Weeks 2, 4, 8, 12
Description: Physician global assessment of all the ways ankylosing spondylitis has affected patient during the last 48 hours. 100 millimeter (mm) Visual Analog Scale (VAS); range: 0=very good to 100=very bad.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF. N = number of subjects with evaluable data.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 42
units on scale
  Week 2 | -15.77 [-21.87 to -9.67] | -7.43 [-13.31 to -1.55]
  Week 4 | -26.25 [-32.35 to -20.15] | -15.23 [-21.11 to -9.35]
  Week 8 | -28.80 [-34.90 to -22.70] | -16.05 [-21.93 to -10.17]
  Week 12 | -32.62 [-38.72 to -26.52] | -17.32 [-23.20 to -11.44]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.054, ANCOVA; Mean Difference (Final Values) = -8.33, 95% CI 2-sided [-16.81 to 0.15] — Least squares mean difference = mean difference final value
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Week 4: Comparison of leasts squares means. Mixed-model analysis of covariance (ANCOVA) using an auto-regressive correlation structure with treatment groups, visits and their interaction as fixed factors, baseline value as a covariate, and patients as a random factor; Test type: Superiority or Other; p = 0.011, ANCOVA; Mean Difference (Final Values) = -11.02, 95% CI [-19.50 to -2.54] — Least squares mean difference = mean difference final value
Statistical Analysis 3: Comparison: Etanercept vs Placebo; Week 8: Comparison of leasts squares means. Mixed-model analysis of covariance (ANCOVA) using an auto-regressive correlation structure with treatment groups, visits and their interaction as fixed factors, baseline value as a covariate, and patients as a random factor; Test type: Superiority or Other; p = 0.003, ANCOVA; Mean Difference (Final Values) = -12.75, 95% CI [-21.23 to -4.27] — Least squares mean difference = mean difference final value
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 15, analysis 3]; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -15.29, 95% CI [-23.7 to -6.82] — Least squares mean difference = mean difference final value

16. Secondary Outcome: Change From Baseline in Physician Global Assessment at Weeks 14, 18, 24
Description: as for outcome 15
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; LOCF.
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
units on scale
  Week 14 | -37.66 [-46.14 to -29.19] | -35.57 [-42.41 to -28.73]
  Week 18 | -43.22 [-49.79 to -36.65] | -37.05 [-44.14 to -29.96]
  Week 24 | -42.68 [-50.25 to -35.10] | -40.41 [-47.64 to -33.17]

17. Secondary Outcome: Normalized Net Incremental Area Under the Curve (AUC) for Nocturnal Back Pain Between Baseline and Week 12
Description: Nocturnal back pain was measured using a 100 millimeter Visual Analog Scale (VAS); range: 0 = none to 100 = extreme. Normalized net incremental area under the curve (AUC) = area between baseline and the Nocturnal Back Pain curve as a function of time (randomization to Week 12); computed using the linear trapezoidal method. All areas above baseline and under the curve are positive and all area below baseline and above the curve are negative. Net incremental AUC = sum of these areas; this result was then divided by the study duration of the patients; negative value = improvement.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF. N=number of subjects with evaluable data.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 41
millimeters | -23.23 [-29.65 to -16.81] | -13.64 [-19.89 to -7.38]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Analysis of covariance (ANCOVA) with treatment as a factor and baseline value as a covariate; Test type: Superiority or Other; p = 0.039, ANCOVA; Mean Difference (Final Values) = -9.59, 95% CI 2-sided [-18.69 to -0.49] — Least squares mean difference = mean difference final value

18. Secondary Outcome: Change From Baseline in Nocturnal Back Pain at Weeks 2, 4, 8, 12
Description: Subject assessment of nocturnal back pain due to ankylosing spondylitis during the last 48 hours using a 100 millimeter (mm) Visual Analog Scale (VAS); range: 0=none to 100=extreme.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
units on scale
  Week 2 | -19.41 [-27.09 to -11.72] | -13.12 [-20.61 to -5.63]
  Week 4 | -20.90 [-28.58 to -13.21] | -15.72 [-23.21 to -8.23]
  Week 8 | -29.27 [-36.95 to -21.58] | -15.54 [-23.03 to -8.05]
  Week 12 | -32.07 [-39.75 to -24.38] | -12.38 [-19.87 to -4.89]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.254, ANCOVA; Mean Difference (Final Values) = -6.28, 95% CI 2-sided [-17.13 to 4.57] — Least squares mean difference = mean difference final value
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.348, ANCOVA; Mean Difference (Final Values) = -5.17, 95% CI [-16.02 to 5.68] — Least squares mean difference = mean difference final value
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 15, analysis 3]; Test type: Superiority or Other; p = 0.014, ANCOVA; Mean Difference (Final Values) = -13.72, 95% CI [-24.57 to -2.88] — Least squares mean difference = mean difference final value
Statistical Analysis 4: Comparison: Etanercept vs Placebo; Week 12: Comparison of leasts squares means. Mixed-model analysis of covariance (ANCOVA) using an auto-regressive correlation structure with treatment groups, visits and their interaction as fixed factors, baseline value as a covariate, and patients as a random factor; Test type: Superiority or Other; p < 0.001, ANCOVA; Mean Difference (Final Values) = -19.69, 95% CI [-30.54 to -8.84] — Least squares mean difference = mean difference final value

19. Secondary Outcome: Change From Baseline in Nocturnal Back Pain at Weeks 14, 18, 24
Description: as for outcome 18
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; LOCF.
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
units on scale
  Week 14 | -36.92 [-46.48 to -27.36] | -27.76 [-37.34 to -18.18]
  Week 18 | -41.73 [-50.58 to -32.87] | -27.89 [-37.91 to -17.86]
  Week 24 | -45.26 [-54.25 to -36.28] | -28.44 [-38.45 to -18.43]

20. Secondary Outcome: Normalized Net Incremental Area Under the Curve (AUC) for Total Back Pain Between Baseline and Week 12
Description: Total back pain was measured using a 100 millimeter Visual Analog Scale (VAS); range: 0 = none to 100 = extreme. Normalized net incremental area under the curve (AUC) = area between baseline and the Total Back Pain curve as a function of time (randomization to Week 12); computed using the linear trapezoidal method. All areas above baseline and under the curve are positive and all area below baseline and above the curve are negative. Net incremental AUC = sum of these areas; this result was then divided by the study duration of the patients; negative value = improvement.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF. N=number of subjects with evaluable data.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 41
millimeters | -21.73 [-28.26 to -15.20] | -13.24 [-19.61 to -6.88]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Analysis of covariance (ANCOVA) with treatment as a factor and baseline value as a covariate; Test type: Superiority or Other; p = 0.071, ANCOVA; Mean Difference (Final Values) = -8.49, 95% CI 2-sided [-17.73 to 0.75] — Least squares mean difference = mean difference final value

21. Secondary Outcome: Change From Baseline in Total Back Pain at Weeks 2, 4, 8, 12
Description: Subject assessment of total back pain due to ankylosing spondylitis during the last 48 hours using a 100 millimeter (mm) Visual Analog Scale (VAS); range: 0=none to 100=extreme.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
units on scale
  Week 2 | -15.37 [-22.99 to -7.76] | -11.80 [-19.22 to -4.38]
  Week 4 | -18.93 [-26.54 to -11.32] | -14.36 [-21.78 to -6.94]
  Week 8 | -28.24 [-35.85 to -20.62] | -15.78 [-23.20 to -8.36]
  Week 12 | -29.18 [-36.79 to -21.57] | -14.93 [-22.35 to -7.51]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.511, ANCOVA; Mean Difference (Final Values) = -3.57, 95% CI 2-sided [-14.31 to 7.17] — Least squares mean difference = mean difference final value
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.401, ANCOVA; Mean Difference (Final Values) = -4.57, 95% CI [-15.31 to 6.17] — Least squares mean difference = mean difference final value
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 15, analysis 3]; Test type: Superiority or Other; p = 0.023, ANCOVA; Mean Difference (Final Values) = -12.45, 95% CI [-23.19 to -1.71] — Least squares mean difference = mean difference final value
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 18, analysis 4]; Test type: Superiority or Other; p = 0.010, ANCOVA; Mean Difference (Final Values) = -14.25, 95% CI [-24.99 to -3.51] — Least squares mean difference = mean difference final value

22. Secondary Outcome: Change From Baseline in Total Back Pain at Weeks 14, 18, 24
Description: Subject assessment of total back pain due to ankylosing spondylitis during the last 48 hours using a 100 millimeter Visual Analog Scale (VAS); range: 0=none to 100=extreme.
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; LOCF.
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
units on scale
  Week 14 | -35.21 [-43.72 to -26.71] | -30.29 [-40.43 to -20.16]
  Week 18 | -40.02 [-48.40 to -31.64] | -31.19 [-42.27 to -20.12]
  Week 24 | -44.50 [-52.74 to -36.25] | -32.27 [-42.71 to -21.83]

23. Secondary Outcome: Normalized Net Incremental Area Under the Curve (AUC) for the Bath Ankylosing Spondylitis Functional Index (BASFI) Between Baseline and Week 12
Description: BASFI was measured using a 100 millimeter Visual Analog Scale (VAS) ranging from 0 = easy to 100 = impossible. Normalized net incremental area under the curve (AUC) = area between baseline and the BASFI curve as a function of time (randomization to Week 12); computed using the linear trapezoidal method. All areas above baseline and under the curve are positive and all area below baseline and above the curve are negative. Net incremental AUC = sum of these areas; this result was then divided by the study duration of the patients; negative value = improvement.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF. N=number of subjects with evaluable data.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 42
millimeters | -14.59 [-19.44 to -9.74] | -9.34 [-14.02 to -4.67]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Analysis of covariance (ANCOVA) with treatment as a factor and baseline as a covariate; Test type: Superiority or Other; p = 0.127, ANCOVA; Mean Difference (Final Values) = -5.25, 95% CI 2-sided [-12.03 to 1.53] — Least squares mean difference = mean difference final value

24. Secondary Outcome: Change From Baseline in the Bath Ankylosing Spondylitis Functional Index (BASFI) at Weeks 2, 4, 8, 12
Description: BASFI is a validated self assessment tool that determines the degree of functional limitation in ankylosing spondylitis (AS) patients using a 100 millimeter (mm) Visual Analog Scale (VAS) measuring level of ability with activities in the last 48 hours; range: 0=easy to 100=impossible. Higher score = greater limitation.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF. N = number of subjects with evaluable data.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 42
units on scale
  Week 2 | -8.23 [-13.82 to -2.63] | -7.80 [-13.19 to -2.41]
  Week 4 | -12.44 [-18.03 to -6.85] | -10.04 [-15.43 to -4.65]
  Week 8 | -19.75 [-25.35 to -14.16] | -11.54 [-16.93 to -6.15]
  Week 12 | -21.63 [-27.22 to -16.03] | -10.09 [-15.47 to -4.70]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.914, ANCOVA; Mean Difference (Final Values) = -0.43, 95% CI 2-sided [-8.23 to 7.38] — Least squares mean difference = mean difference final value
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.544, ANCOVA; Mean Difference (Final Values) = -2.40, 95% CI [-10.21 to 5.41] — Least squares mean difference = mean difference final value
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 15, analysis 3]; Test type: Superiority or Other; p = 0.039, ANCOVA; Mean Difference (Final Values) = -8.21, 95% CI [-16.02 to -0.40] — Least squares mean difference = mean difference final value
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 18, analysis 4]; Test type: Superiority or Other; p = 0.004, ANCOVA; Mean Difference (Final Values) = -11.54, 95% CI [-19.35 to -3.73] — Least squares mean difference = mean difference final value

25. Secondary Outcome: Bath Ankylosing Functional Index (BASFI): Independent Components at Weeks 2, 4, 8, 12
Description: Subject rating of last 48 hours, 100 millimeter Visual Analog Scale; range 0=easy to 100=impossible: 1)Putting on socks/tights without (w/o) help; 2)Bending forward from waist to pickup pen from floor w/o aid; 3)Reaching to high shelf w/o aid; 4)Getting out of armless dining room chair w/o using hands/other help; 5)Getting up off floor w/o help from lying on back; 6)Standing unsupported 10 minutes w/o discomfort; 7)Climbing 12-15 steps w/o handrail or walking aid; 8)Looking over shoulder w/o turning body; 9) Doing physically demanding activities; 10) Doing full days activities (home or work).
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; in the case of missing data, no replacement or imputation method was performed. Abbreviations: C = component (number), Act = Activities.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
units on a scale
  Baseline C1: Putting on Socks or Tights | 51.1 [42.8 to 59.4] | 43.8 [35.7 to 52.0]
  Week 2 C1: Putting on Socks or Tights | 47.6 [37.9 to 57.3] | 36.5 [27.4 to 45.5]
  Week 4 C1: Putting on Socks or Tights | 41.1 [31.4 to 50.8] | 32.7 [24.0 to 41.4]
  Week 8 C1: Putting on Socks or Tights | 32.3 [24.0 to 40.7] | 30.6 [22.0 to 39.1]
  Week 12 C1: Putting on Socks or Tights | 33.2 [23.4 to 43.0] | 36.0 [24.6 to 45.6]
  Baseline C2: Bending from Waist | 63.4 [54.2 to 72.7] | 61.5 [52.6 to 70.5]
  Week 2 C2: Bending from Waist | 54.1 [43.0 to 65.3] | 55.7 [45.5 to 65.9]
  Week 4 C2: Bending from Waist | 51.1 [39.1 to 63.0] | 54.0 [44.1 to 63.9]
  Week 8 C2: Bending from Waist | 43.3 [32.3 to 54.3] | 54.2 [43.5 to 64.9]
  Week 12 C2: Bending from Waist | 41.1 [29.8 to 52.4] | 56.2 [45.6 to 66.7]
  Baseline C3: Reaching to High Shelf | 61.5 [52.5 to 70.6] | 54.3 [46.3 to 62.3]
  Week 2 C3: Reaching to High Shelf | 52.1 [41.9 to 62.2] | 50.3 [40.8 to 59.7]
  Week 4 C3: Reaching to High Shelf | 50.2 [39.7 to 60.7] | 43.8 [35.2 to 52.4]
  Week 8 C3: Reaching to High Shelf | 37.4 [27.7 to 47.1] | 44.1 [36.4 to 51.8]
  Week 12 C3: Reaching to High Shelf | 37.3 [26.8 to 47.9] | 44.5 [36.2 to 52.8]
  Baseline C4: Getting Out Armless Chair | 55.8 [46.1 to 65.5] | 47.5 [38.8 to 56.2]
  Week 2 C4: Getting Out Armless Chair | 47.2 [36.7 to 57.6] | 38.1 [29.0 to 47.2]
  Week 4 C4: Getting Out Armless Chair | 42.1 [31.0 to 53.3] | 36.1 [27.7 to 44.6]
  Week 8 C4: Getting Out Armless Chair | 33.6 [24.3 to 42.9] | 35.1 [25.9 to 44.3]
  Week 12 C4: Getting Out Armless Chair | 31.7 [21.7 to 41.7] | 36.5 [26.8 to 46.3]
  Baseline C5: Getting Up Off Floor | 71.8 [64.1 to 79.5] | 60.8 [52.7 to 68.9]
  Week 2 C5: Getting Up Off Floor | 57.0 [46.7 to 67.3] | 49.4 [40.1 to 58.8]
  Week 4 C5: Getting Up Off Floor | 55.0 [44.5 to 65.6] | 48.5 [39.4 to 57.5]
  Week 8 C5: Getting Up Off Floor | 43.7 [32.9 to 54.4] | 44.2 [34.7 to 53.7]
  Week 12 C5: Getting Up Off Floor | 44.5 [33.7 to 55.2] | 46.1 [36.7 to 55.5]
  Baseline C6: Standing Unsupported | 58.9 [49.9 to 67.9] | 49.0 [39.7 to 58.3]
  Week 2 C6: Standing Unsupported | 50.8 [40.4 to 61.2] | 44.9 [35.5 to 54.3]
  Week 4 C6: Standing Unsupported | 46.4 [35.8 to 57.0] | 42.0 [33.6 to 50.3]
  Week 8 C6: Standing Unsupported | 40.8 [30.9 to 50.7] | 40.9 [31.6 to 50.1]
  Week 12 C6: Standing Unsupported | 39.0 [28.3 to 49.7] | 42.2 [32.5 to 51.9]
  Baseline C7: Climbing 12-15 Steps | 55.0 [45.3 to 64.8] | 47.5 [37.9 to 57.1]
  Week 2 C7: Climbing 12-15 Steps | 47.4 [36.7 to 58.1] | 38.4 [29.3 to 47.4]
  Week 4 C7: Climbing 12-15 Steps | 42.3 [31.8 to 52.8] | 37.4 [28.4 to 46.4]
  Week 8 C7: Climbing 12-15 Steps | 37.4 [27.5 to 47.3] | 35.6 [25.8 to 45.3]
  Week 12 C7: Climbing 12-15 Steps | 35.0 [24.7 to 45.2] | 32.9 [23.6 to 42.3]
  Baseline C8: Looking Over Shoulder | 81.0 [74.0 to 87.9] | 81.9 [75.7 to 88.0]
  Week 2 C8: Looking Over Shoulder | 72.9 [64.3 to 81.5] | 68.4 [59.5 to 77.2]
  Week 4 C8: Looking Over Shoulder | 63.7 [53.5 to 74.0] | 71.6 [62.8 to 80.4]
  Week 8 C8: Looking Over Shoulder | 56.9 [45.9 to 67.9] | 71.1 [61.6 to 80.7]
  Week 12: C8: Looking Over Shoulder | 54.1 [43.0 to 65.2] | 68.1 [58.8 to 77.4]
  Baseline C9: Physically Demanding Act | 67.6 [60.7 to 74.5] | 65.4 [59.2 to 71.6]
  Week 2 C9: Physically Demanding Act | 60.7 [51.7 to 69.6] | 58.4 [51.4 to 65.4]
  Week 4 C9: Physically Demanding Act | 53.0 [43.4 to 62.6] | 53.6 [46.4 to 60.8]
  Week 8 C9: Physically Demanding Act | 48.4 [38.4 to 58.3] | 47.8 [40.5 to 55.1]
  Week 12 C9: Physically Demanding Act | 43.2 [33.4 to 52.9] | 54.9 [47.7 to 62.1]
  Baseline C10: Full Days Act | 66.9 [59.4 to 74.5] | 57.1 [49.4 to 64.8]
  Week 2 C10: Full Days Act | 57.2 [48.7 to 65.7] | 49.3 [42.1 to 56.5]
  Week 4 C10: Full Days Act | 52.4 [43.3 to 61.4] | 51.6 [43.7 to 59.5]
  Week 8 C10: Full Days Act | 47.6 [37.3 to 57.8] | 44.4 [37.5 to 51.3]
  Week 12 C10: Full Days Act | 43.1 [32.2 to 53.9] | 49.0 [40.9 to 57.2]

26. Secondary Outcome: Bath Ankylosing Functional Index (BASFI) Independent Components at Weeks 14, 18, 24
Description: Subject rating of last 48 hours, 100 mm Visual Analog Scale; range 0=easy to 100=impossible: 1) Putting on socks/tights without (w/o) help; 2) Bending forward from waist to pickup pen from floor w/o aid; 3) Reaching to high shelf w/o aid; 4) Getting out of armless dining room chair w/o using hands/other help; 5) Getting up off floor w/o help from lying on back; 6) Standing unsupported 10 minutes w/o discomfort; 7) Climbing 12-15 steps w/o handrail or walking aid; 8) Looking over shoulder w/o turning body; 9) Doing physically demanding activities; 10) Doing full days activities (home or work).
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; in the case of missing data, no replacement or imputation method was performed. Abbreviations: C=component (number), Act=Activities.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
units on a scale
  Week 14 C1: Putting on Socks or Tights | 32.7 [22.6 to 42.8] | 25.7 [16.6 to 34.8]
  Week 18 C1: Putting on Socks or Tights | 31.3 [21.3 to 41.2] | 26.6 [17.1 to 36.1]
  Week 24 C1: Putting on Socks or Tights | 26.7 [16.8 to 36.5] | 24.5 [15.4 to 33.6]
  Week 14 C2: Bending from Waist | 42.1 [29.6 to 54.6] | 47.1 [35.9 to 58.4]
  Week 18 C2: Bending from Waist | 36.9 [25.0 to 48.8] | 45.3 [32.9 to 57.7]
  Week 24 C2: Bending from Waist | 36.1 [23.9 to 48.3] | 44.6 [33.0 to 56.3]
  Week 14 C3: Reaching to High Shelf | 37.0 [26.0 to 48.0] | 31.7 [22.8 to 40.6]
  Week 18 C3: Reaching to High Shelf | 32.1 [21.7 to 42.6] | 34.2 [25.0 to 43.5]
  Week 24 C3: Reaching to High Shelf | 27.4 [18.1 to 36.7] | 32.1 [23.8 to 40.4]
  Week 14 C4: Getting Out Armless Chair | 32.0 [20.9 to 43.2] | 27.9 [18.3 to 37.6]
  Week 18 C4: Getting Out Armless Chair | 27.3 [17.2 to 37.4] | 26.5 [16.9 to 36.1]
  Week 24 C4: Getting Out Armless Chair | 23.4 [14.6 to 32.3] | 26.2 [17.1 to 35.3]
  Week 14 C5: Getting Up Off Floor | 43.6 [31.1 to 56.1] | 36.3 [26.6 to 46.1]
  Week 18 C5: Getting Up Off Floor | 40.0 [28.1 to 51.8] | 36.5 [26.6 to 46.3]
  Week 24 C5: Getting Up Off Floor | 38.2 [27.0 to 49.4] | 34.4 [24.1 to 44.7]
  Week 14 C6: Standing Unsupported | 38.8 [27.2 to 50.3] | 29.7 [20.8 to 38.6]
  Week 18 C6: Standing Unsupported | 32.6 [22.1 to 43.2] | 33.3 [22.9 to 43.7]
  Week 24 C6: Standing Unsupported | 30.5 [20.7 to 40.3] | 33.8 [24.1 to 43.6]
  Week 14 C7: Climbing 12-15 Steps | 34.0 [22.4 to 45.6] | 26.7 [17.7 to 35.7]
  Week 18 C7: Climbing 12-15 Steps | 30.7 [20.0 to 41.3] | 27.4 [17.2 to 37.6]
  Week 24 C7: Climbing 12-15 Steps | 28.8 [18.7 to 38.9] | 27.1 [17.0 to 37.2]
  Week 14 C8: Looking Over Shoulder | 52.4 [40.2 to 64.5] | 58.6 [47.5 to 69.8]
  Week 18 C8: Looking Over Shoulder | 50.7 [38.6 to 62.7] | 57.7 [46.9 to 68.5]
  Week 24 C8: Looking Over Shoulder | 46.4 [34.2 to 58.6] | 55.3 [44.8 to 65.9]
  Week 14 C9: Physically Demanding Act | 41.8 [30.7 to 53.0] | 37.3 [29.9 to 44.7]
  Week 18 C9: Physically Demanding Act | 38.6 [28.5 to 48.8] | 43.5 [34.9 to 52.1]
  Week 24 C9: Physically Demanding Act | 33.7 [23.7 to 43.6] | 38.5 [29.9 to 47.1]
  Week 14 C10: Full Days Act | 40.4 [29.2 to 51.6] | 36.1 [27.7 to 44.4]
  Week 18 C10: Full Days Act | 37.9 [26.7 to 49.0] | 40.0 [30.9 to 49.0]
  Week 24 C10: Full Days Act | 32.1 [22.6 to 41.6] | 37.5 [28.4 to 46.5]

27. Secondary Outcome: Change From Baseline in the Bath Ankylosing Spondylitis Disease Activity Index (BASDAI) at Weeks 2, 4, 8, 12
Description: BASDAI is a validated self assessment tool used to determine disease activity in patients with ankylosing spondylitis in the last 48 hours. Utilizing a Visual Analog Scale (VAS) of 0-10 (0=none and 10=very severe) patient's answered 6 questions measuring discomfort, pain and fatigue. The BASDAI final mean score was calculated taking all 6 VAS assessments.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
units on a scale
  Week 2 | -14.25 [-20.51 to -7.99] | -7.39 [-13.34 to -1.43]
  Week 4 | -18.41 [-24.67 to -12.15] | -11.97 [-17.92 to -6.01]
  Week 8 | -26.06 [-32.31 to -19.80] | -13.51 [-19.46 to -7.55]
  Week 12 | -26.38 [-32.64 to -20.12] | -14.43 [-20.39 to -8.47]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.122, ANCOVA; Mean Difference (Final Values) = -6.86, 95% CI 2-sided [-15.57 to 1.85] — Least squares mean difference = mean difference final value
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.145, ANCOVA; Mean Difference (Final Values) = -6.45, 95% CI [-15.16 to 2.26] — Least squares mean difference = mean difference final value
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 15, analysis 3]; Test type: Superiority or Other; p = 0.005, ANCOVA; Mean Difference (Final Values) = -12.55, 95% CI [-21.26 to -3.84] — Least squares mean difference = mean difference final value
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 18, analysis 4]; Test type: Superiority or Other; p = 0.008, ANCOVA; Mean Difference (Final Values) = -11.95, 95% CI [-20.66 to -3.24] — Least squares mean difference = mean difference final value

28. Secondary Outcome: Change From Baseline in the Bath Ankylosing Spondylitis (AS) Disease Activity Index (BASDAI) at Weeks 14, 18, 24
Description: BASDAI is a validated self assessment tool used to determine disease activity in patients with ankylosing spondylitis (AS) in the last 48 hours. Utilizing a Visual Analog Scale (VAS) of 0-10 (0=none and 10=very severe) patient's answered 6 questions measuring discomfort, pain and fatigue. The BASDAI final mean score was calculated taking all 6 VAS assessments.
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; LOCF.
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
units on scale
  Week 14 | -29.26 [-37.34 to -21.17] | -27.41 [-34.52 to -20.30]
  Week 18 | -34.20 [-41.89 to -26.52] | -28.21 [-35.94 to -20.47]
  Week 24 | -37.62 [-44.97 to -30.27] | -28.62 [-36.49 to -20.76]

29. Secondary Outcome: Bath Ankylosing Spondylitis (AS) Disease Activity Index (BASDAI) Independent Components at Weeks 2, 4, 8, 12
Description: BASDAI subject rated components over last 48 hours using 100 mm Visual Analog Scale; components 1-5: range 0=none to 100=very severe; component 6: range:0=0 hours to 100=2 hours or more. 1) Overall level of fatigue/tiredness experienced; 2) Overall level of AS neck,back or hip pain experienced; 3) Overall level of pain/swelling in joints other than neck, back or hips; 4) Overall level of discomfort from any areas tender to touch or pressure; 5) Overall level of morning stiffness from time of awakening; 6) Duration of morning stiffness from time of awakening, and morning stiffness subscale.
Time Frame: Week 2, Week 4, Week 8, Week 12
Population: mITT; in case of mising data, no replacement or imputation method was performed. Abbreviations: C=component, AS=Ankylosing Spondylitis.
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
units on scale
  Baseline C1: Fatigue/Tiredness | 68.2 [62.5 to 73.8] | 61.9 [57.1 to 66.8]
  Week 2 C1: Fatigue/Tiredness | 56.6 [48.7 to 64.5] | 55.8 [49.1 to 62.5]
  Week 4 C1: Fatigue/Tiredness | 51.4 [43.1 to 59.6] | 54.2 [47.0 to 61.4]
  Week 8 C1: Fatigue/Tiredness | 44.4 [36.2 to 52.7] | 50.9 [43.3 to 58.5]
  Week 12 C1: Fatigue/Tiredness | 43.9 [33.9 to 53.9] | 48.5 [40.1 to 56.9]
  Baseline C2: AS Neck, Back or Hip Pain | 73.0 [68.7 to 77.3] | 68.1 [63.4 to 72.9]
  Week 2 C2: AS Neck, Back or Hip Pain | 53.9 [45.7 to 62.1] | 57.6 [50.2 to 65.0]
  Week 4 C2: AS Neck, Back or Hip Pain | 51.5 [43.0 to 60.0] | 55.0 [47.2 to 62.9]
  Week 8 C2: AS Neck, Back or Hip Pain | 41.4 [32.8 to 50.1] | 52.1 [45.0 to 59.2]
  Week 12 C2: AS Neck, Back or Hip Pain | 41.0 [31.8 to 50.2] | 52.0 [44.5 to 59.5]
  Baseline C3: Pain/Swelling in Other Joints | 49.3 [41.1 to 57.5] | 45.3 [36.1 to 54.4]
  Week 2 C3: Pain/Swelling in Other Joints | 39.2 [29.5 to 48.9] | 41.7 [31.7 to 51.7]
  Week 4 C3: Pain/Swelling in Other Joints | 37.3 [27.8 to 46.8] | 38.2 [30.0 to 46.5]
  Week 8 C3: Pain/Swelling in Other Joints | 30.1 [20.8 to 39.5] | 40.4 [32.0 to 48.8]
  Week 12 C3: Pain/Swelling in Other Joints | 31.8 [21.7 to 41.8] | 37.9 [29.6 to 46.2]
  Baseline C4: Discomfort Areas Tender to Touch | 62.3 [55.5 to 69.2] | 57.2 [49.9 to 64.4]
  Week 2 C4: Discomfort Areas Tender to Touch | 42.1 [32.5 to 51.6] | 51.9 [43.3 to 60.4]
  Week 4 C4: Discomfort Areas Tender to Touch | 38.3 [29.0 to 47.5] | 41.5 [33.2 to 49.9]
  Week 8 C4: Discomfort Areas Tender to Touch | 31.2 [22.6 to 39.9] | 40.7 [32.5 to 48.8]
  Week 12 C4: Discomfort Areas Tender to Touch | 28.8 [19.9 to 37.7] | 38.0 [30.5 to 45.4]
  Baseline C5: Morning Stiffness | 70.8 [64.8 to 76.8] | 66.3 [61.6 to 70.9]
  Week 2 C5: Morning Stiffness | 51.3 [42.9 to 59.8] | 55.6 [48.7 to 62.4]
  Week 4 C5: Morning Stiffness | 46.5 [37.2 to 55.7] | 50.7 [43.6 to 57.8]
  Week 8 C5: Morning Stiffness | 38.1 [29.1 to 47.2] | 44.7 [37.4 to 52.0]
  Week 12 C5: Morning Stiffness | 37.8 [27.6 to 48.1] | 44.8 [37.7 to 52.0]
  Baseline C6: Duration Morning Stiffness | 62.1 [53.9 to 70.3] | 52.4 [44.5 to 60.3]
  Week 2 C6: Duration Morning Stiffness | 46.8 [36.6 to 57.0] | 44.0 [35.7 to 52.3]
  Week 4 C6: Duration Morning Stiffness | 42.2 [31.9 to 52.6] | 43.0 [35.2 to 50.9]
  Week 8 C6: Duration Morning Stiffness | 34.6 [24.2 to 44.9] | 43.7 [36.1 to 51.4]
  Week 12 C6: Duration Morning Stiffness | 34.9 [24.0 to 45.8] | 44.7 [36.1 to 53.3]
  Baseline: Subscore Morning Stiffness (n=39, 43) | 66.45 [60.42 to 72.48] | 59.34 [54.19 to 64.48]
  Week 2: Subscore Morning Stiffness | 49.72 [41.16 to 58.29] | 49.78 [42.88 to 56.68]
  Week 4: Subscore Morning Stiffness | 44.34 [35.58 to 53.11] | 46.87 [39.83 to 53.91]
  Week 8: Subscore Morning Stiffness | 36.34 [27.19 to 45.48] | 44.22 [37.20 to 51.24]
  Week 12: Subscore Morning Stiffness | 36.39 [26.41 to 46.37] | 44.77 [37.41 to 52.13]

30. Secondary Outcome: Bath Ankylosing Spondylitis (AS) Disease Activity Index (BASDAI) Independent Components at Weeks 14, 18, 24
Description: BASDAI subject rated components over last 48 hours using a 100 millimeter Visual Analog Scale; components 1-5: range 0=none to 100=very severe; component 6: range:0=0 hours to 100=2 hours or more. 1) Overall level of fatigue/tiredness experienced; 2) Overall level of AS neck,back or hip pain experienced; 3)Overall level of pain/swelling in joints other than neck,back or hips; 4) Overall level of discomfort from any areas tender to touch or pressure; 5) Overall level of morning stiffness from time of awakening; 6) Duration of morning stiffness from time of awakening.
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; in case of missing data, no replacement or imputation method was performed. Abbreviations: C=component, AS=Ankylosing Spondylitis.
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
units on scale
  Week 14 C1: Fatigue/Tiredness | 41.7 [31.4 to 52.0] | 38.3 [29.5 to 47.0]
  Week 18 C1: Fatigue/Tiredness | 33.1 [24.0 to 42.2] | 38.9 [28.9 to 48.9]
  Week 24 C1: Fatigue/Tiredness | 28.0 [20.1 to 35.9] | 35.3 [25.5 to 45.1]
  Week 14 C2: AS Neck, Back or Hip Pain | 39.9 [29.6 to 50.1] | 35.0 [26.8 to 43.3]
  Week 18 C2: AS Neck, Back or Hip Pain | 35.1 [26.2 to 44.0] | 35.0 [25.7 to 44.3]
  Week 24 C2: AS Neck, Back or Hip Pain | 28.2 [19.5 to 36.8] | 30.0 [21.3 to 38.7]
  Week 14 C3: Pain/Swelling in Other Joints | 27.0 [17.3 to 36.8] | 28.4 [20.5 to 36.3]
  Week 18 C3: Pain/Swelling in Other Joints | 23.8 [14.5 to 33.1] | 26.4 [17.4 to 35.4]
  Week 24 C3: Pain/Swelling in Other Joints | 21.0 [12.5 to 29.4] | 24.9 [16.5 to 33.3]
  Week 14 C4: Discomfort Areas Tender to Touch | 30.0 [19.9 to 40.0] | 29.1 [21.2 to 36.9]
  Week 18 C4: Discomfort Areas Tender to Touch | 24.1 [15.4 to 32.8] | 28.7 [19.6 to 37.9]
  Week 24 C4: Discomfort Areas Tender to Touch | 19.3 [11.9 to 26.8] | 25.6 [17.5 to 33.8]
  Week 14 C5: Morning Stiffness | 35.8 [25.6 to 46.1] | 28.5 [20.3 to 36.7]
  Week 18 C5: Morning Stiffness | 31.4 [21.5 to 41.4] | 28.6 [20.2 to 37.0]
  Week 24 C5: Morning Stiffness | 26.4 [17.5 to 35.4] | 24.7 [17.8 to 31.7]
  Week 14 C6: Duration Morning Stiffness | 31.3 [20.9 to 41.6] | 27.7 [19.4 to 36.0]
  Week 18 C6: Duration Morning Stiffness | 31.3 [20.9 to 41.7] | 25.7 [17.6 to 33.9]
  Week 24 C6: Duration Morning Stiffness | 24.9 [15.4 to 34.4] | 24.4 [17.2 to 31.6]
  Week 14: Subscore Morning Stiffness | 33.5 [24.03 to 43.06] | 28.09 [20.14 to 36.04]
  Week 18: Subscore Morning Stiffness | 31.38 [21.66 to 41.10] | 27.17 [19.02 to 35.32]
  Week 24: Subscore Morning Stiffness | 25.40 [16.69 to 34.12] | 24.55 [17.77 to 31.34]

31. Secondary Outcome: Normalized Net Incremental Area Under the Curve (AUC) for Bath Ankylosing Spondylitis-Global Score (BAS-G) Visual Analog Scale Between Baseline and Week 12
Description: BAS-G was measured using a 100 millimeter Visual Analog Scale (VAS) ranging from 0=none to 100=very important. Normalized net incremental area under the curve (AUC) = area between baseline and the BAS-G curve as a function of time (randomization to Week 12); computed using the linear trapezoidal method. All areas above baseline and under the curve are positive and all area below baseline and above the curve are negative. Net incremental AUC = sum of these areas; this result was then divided by the study duration of the patients; negative value = improvement.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF. N=number of subjects with evaluable data.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 38 | 42
millimeters | -21.36 [-27.07 to -15.66] | -15.43 [-20.85 to -10.00]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Analysis of covariance (ANCOVA) with treatment as a factor and baseline value as a covariate; Test type: Superiority or Other; p = 0.139, ANCOVA; Mean Difference (Final Values) = -5.94, 95% CI 2-sided [-13.84 to 1.96] — Least squares mean difference = mean difference final value

32. Secondary Outcome: Change From Baseline in the Bath Ankylosing Spondylitis-Global Score (BAS-G) at Weeks 2, 4, 8, 12
Description: Subject assessment of the effect of their disease on well-being over last 48 hours using a 100 millimeter (mm) Visual Analog Scale (VAS); range: 0=none to 100=very important.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF. N=number of subjects with evaluable data.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 38 | 42
units on scale
  Week 2 | -13.74 [-20.81 to -6.68] | -14.64 [-21.36 to -7.92]
  Week 4 | -20.09 [-27.16 to -13.02] | -14.99 [-21.71 to -8.27]
  Week 8 | -28.17 [-35.24 to -21.11] | -18.27 [-24.99 to -11.55]
  Week 12 | -29.78 [-36.84 to -22.71] | -16.12 [-22.84 to -9.40]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 12, analysis 1]; Test type: Superiority or Other; p = 0.857, ANCOVA; Mean Difference (Final Values) = 0.89, 95% CI 2-sided [-8.88 to 10.67] — Least squares mean difference = mean difference final value
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 15, analysis 2]; Test type: Superiority or Other; p = 0.304, ANCOVA; Mean Difference (Final Values) = -5.10, 95% CI [-14.88 to 4.67] — Least squares mean difference = mean difference final value
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 15, analysis 3]; Test type: Superiority or Other; p = 0.047, ANCOVA; Mean Difference (Final Values) = -9.90, 95% CI [-19.68 to -0.13] — Least squares mean difference = mean difference final value
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 18, analysis 4]; Test type: Superiority or Other; p = 0.007, ANCOVA; Mean Difference (Final Values) = -13.65, 95% CI [-23.43 to -3.88] — Least squares mean difference = mean difference final value

33. Secondary Outcome: Change From Baseline in the Bath Ankylosing Spondylitis-Global Score (BAS-G) at Weeks 14, 18, 24
Description: Subject assessment of the effect of their disease on well-being over last 48 hours using a 100 millimeter Visual Analog Scale (VAS); range: 0=none to 100=very important.
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; LOCF.
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
units on scale
  Week 14 | -34.29 [-43.58 to -25.00] | -34.93 [-44.51 to -25.34]
  Week 18 | -36.93 [-45.27 to -28.60] | -35.98 [-44.69 to -27.26]
  Week 24 | -42.35 [-50.58 to -34.13] | -35.89 [-44.30 to -27.48]

34. Secondary Outcome: Bath Ankylosing Spondylitis Global Score (BAS-G) Independent Component: Effect of Disease on Well-being at Weeks 2, 4, 8, 12
Description: Subject evaluation of the effect of their disease on well-being over the last week using a using a 100 millimeter Visual Anaog Scale; range: 0=none to 100=very important.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF.
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
units on scale
  Baseline | 72.1 [66.9 to 77.4] | 68.3 [62.6 to 73.9]
  Week 2 | 57.8 [49.9 to 65.6] | 54.4 [47.4 to 61.4]
  Week 4 | 51.4 [43.5 to 59.4] | 54.0 [46.8 to 61.3]
  Week 8 | 43.3 [34.9 to 51.6] | 50.8 [44.9 to 56.7]
  Week 12 | 42.1 [33.0 to 51.1] | 52.9 [46.3 to 59.5]

35. Secondary Outcome: Change From Baseline to Week 12 in Forced Vital Capacity (FVC), Vital Capacity (VC), and Forced Expiratory Volume in One Second (FEV1)
Time Frame: Baseline, Week 12
Population: mITT. In the case of missing data, no replacement or imputation method was performed.
Measure: Least Squares Mean (95% Confidence Interval); unit: liters
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
liters
  Vital Capacity | 0.14 [0.05 to 0.23] | -0.05 [-0.14 to 0.04]
  Forced Vital Capacity (FVC) | 0.16 [0.07 to 0.25] | -0.02 [-0.11 to 0.07]
  Forced Expiratory Volume in 1 Second | 0.05 [-0.02 to 0.12] | -0.02 [-0.09 to 0.05]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Vital Capacity: Analysis of covariance (ANCOVA) with treatment as a factor and baseline value as a covariate; Test type: Superiority or Other; p = 0.003, ANCOVA; Mean Difference (Final Values) = 0.19, 95% CI 2-sided [0.06 to 0.31] — Least squares mean difference = mean difference final value
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Forced Vital Capacity: Analysis of covariance (ANCOVA) with treatment as a factor and baseline value as a covariate; Test type: Superiority or Other; p = 0.006, ANCOVA; Mean Difference (Final Values) = 0.18, 95% CI 2-sided [0.05 to 0.31] — Least squares mean difference = mean difference final value
Statistical Analysis 3: Comparison: Etanercept vs Placebo; Forced Expitatory Volume in 1 second: Analysis of covariance (ANCOVA) with treatment as a factor and baseline value as a covariate; Test type: Superiority or Other; p = 0.205, ANCOVA; Mean Difference (Final Values) = 0.06, 95% CI 2-sided [-0.04 to 0.17] — Least squares mean difference = mean difference final value

36. Secondary Outcome: Change From Baseline to Week 12 in Ratio Forced Expitatory Volume in One Second (FEV1)/Forced Vital Capacity (FVC) (%)
Time Frame: Baseline, Week 12
Population: mITT; N=number of subjects with evaluable data. In the case of missing data, no replacement or imputation method was performed.
Measure: Least Squares Mean (95% Confidence Interval); unit: percent
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 37 | 38
percent | -2.49 [-4.15 to -0.84] | 0.10 [-1.53 to 1.73]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Analysis oaf covariance (ANCOVA) with treatment as a factor and baseline value as a covariate; Test type: Superiority or Other; p = 0.030, ANCOVA; Mean Difference (Final Values) = -2.59, 95% CI 2-sided [-4.93 to -0.26] — Least squares mean difference = mean difference final value

37. Secondary Outcome: Normalized Net Incremental Area Under the Curve (AUC) for the Bath Ankylosing Spondylitis Metrology Index (BASMI) Between Baseline and Week 12
Description: BASMI was composed of 5 measures; each measure scored 0-2 (0=normal mobility, 2=severe reduction); final score range: 0 to 10. Normalized net incremental area under the curve (AUC) = area between baseline and the BASMI curve as a function of time (randomization to Week 12); computed using the linear trapezoidal method. All areas above baseline and under the curve are positive and all area below baseline and above the curve are negative. Net incremental AUC = sum of these areas; this result was then divided by the study duration of the patients; negative value = improvement.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
millimeters | -0.41 [-0.57 to -0.26] | -0.18 [-0.33 to -0.03]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Analysis of covariance (ANCOVA) with treatment as a factor and baseline value as covariate; Test type: Superiority or Other; p = 0.035, ANCOVA; Mean Difference (Final Values) = -0.23, 95% CI 2-sided [-0.45 to -0.02] — Least squares mean difference = mean difference final value

38. Secondary Outcome: Change From Baseline in Spinal Mobility Measured With the Bath Ankylosing Spondylitis Metrology Index (BASMI) at Weeks 2, 4, 8, 12
Description: BASMI is an objective measure of spinal mobility. The BASMI score is composed of 5 measures: cervical rotation, intermalleolar distance, modified Schober test, lateral flexion and tragus to wall distance. Each measure was scored 0-2 (0=normal mobility, 2=severe reduction) to give a final score ranging 0 to 10. Higher score = greater reduction in spinal mobility.
Time Frame: Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
units on scale
  Week 2 | -0.27 [-0.47 to -0.06] | -0.17 [-0.37 to 0.02]
  Week 4 | -0.37 [-0.58 to -0.17] | -0.23 [-0.43 to -0.04]
  Week 8 | -0.57 [-0.77 to -0.36] | -0.18 [-0.38 to 0.01]
  Week 12 | -0.57 [-0.77 to -0.36] | -0.20 [-0.40 to -0.01]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Week 2: Mixed model analysis of covariance (ANCOVA), using an auto-regressive correlation structure, with treatment groups, visits and their interaction as fixed factors, baseline value as a covariate and patients as a random factor; Test type: Superiority or Other; p = 0.515, ANCOVA; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.38 to 0.19] — Least squares mean difference = mean difference final value
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Week 4: Mixed model analysis of covariance (ANCOVA), using an auto-regressive correlation structure, with treatment groups, visits and their interaction as fixed factors, baseline value as a covariate and patients as a random factor; Test type: Superiority or Other; p = 0.316, ANCOVA; Mean Difference (Final Values) = -0.14, 95% CI [-0.43 to 0.14] — Least squares mean difference = mean difference final value
Statistical Analysis 3: Comparison: Etanercept vs Placebo; Week 8: Mixed model analysis of covariance (ANCOVA), using an auto-regressive correlation structure, with treatment groups, visits and their interaction as fixed factors, baseline value as a covariate and patients as a random factor; Test type: Superiority or Other; p = 0.008, ANCOVA; Mean Difference (Final Values) = -0.39, 95% CI [-0.67 to -0.10] — Least squares mean difference = mean difference final value
Statistical Analysis 4: Comparison: Etanercept vs Placebo; Week 12: Mixed model analysis of covariance (ANCOVA), using an auto-regressive correlation structure, with treatment groups, visits and their interaction as fixed factors, baseline value as a covariate and patients as a random factor; Test type: Superiority or Other; p = 0.011, ANCOVA; Mean Difference (Final Values) = -0.37, 95% CI [-0.65 to -0.08] — Least squares mean difference = mean difference final value

39. Secondary Outcome: Change From Baseline in Spinal Mobility Measured With the Bath Ankylosing Spondylitis Metrology Index (BASMI) at Weeks 14, 18, 24
Description: BASMI is an objective measure of spinal mobility. The BASMI score is composed of 5 measures: cervical rotation, intermalleolar distance, modified Schober's test, lateral flexion and tragus to wall distance. Each measure was scored 0-2 (0=normal mobility, 2=severe reduction) to give a final score ranging 0 to 10. Higher score = greater reduction in spinal mobility.
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; LOCF.
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
units on scale
  Week 14 | -0.73 [-0.98 to -0.49] | -0.49 [-0.68 to -0.30]
  Week 18 | -0.65 [-0.94 to -0.36] | -0.49 [-0.69 to -0.29]
  Week 24 | -0.80 [-1.05 to -0.55] | -0.50 [-0.72 to -0.29]

40. Secondary Outcome: Bath Ankylosing Spondylitis Metrology Index (BASMI) Independent Component: Cervical Rotation at Weeks 2, 4, 8, 12
Description: Cervical rotation: measurement of degrees to which the subjects could turn their heads as far as possible to the right and then to the left. Mean of ordinal scores from 0: >= 85 degrees to 10: <= 8.5 degrees.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF. In the case of missing data, no replacement or imputation method was performed.
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
units on scale
  Baseline | 39.85 [33.77 to 45.92] | 37.14 [30.37 to 43.91]
  Week 2 | 43.05 [35.73 to 50.38] | 38.34 [32.08 to 44.60]
  Week 4 | 42.55 [35.64 to 49.47] | 39.67 [33.21 to 46.14]
  Week 8 | 44.34 [37.57 to 51.11] | 39.79 [32.44 to 47.14]
  Week 12 | 46.39 [39.55 to 53.24] | 42.67 [35.58 to 49.75]

41. Secondary Outcome: Bath Ankylosing Spondylitis Metrology Index (BASMI): Spinal Mobility Measured With Cervical Rotation at Weeks 14, 18, 24
Description: Cervical rotation: measurement in degree to which the subjects could turn their heads as far as possible to the right and then to the left. Mean of ordinal scores from 0: >= 85 degrees to 10: <= 8.5 degrees.
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; in the case of missing data, no replacement or imputation method was performed.
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
units on scale
  Week 14 | 47.75 [40.85 to 54.65] | 44.78 [37.32 to 52.24]
  Week 18 | 44.62 [37.20 to 52.03] | 43.92 [36.57 to 51.27]
  Week 24 | 48.74 [41.78 to 55.71] | 43.82 [36.26 to 51.37]

42. Secondary Outcome: Bath Ankylosing Spondylitis Metrology Index (BASMI) Independent Component: Spinal Mobility Measured With Tragus-to-wall Distance at Baseline and Weeks 2, 4, 8, 12
Description: Measurement in centimeters (cm) of distance between the tragus and wall from right and left side while subject is standing with back against the wall; knees straight; scapulae, buttocks, and heels against the wall; with head in neutral position. Measurement of two attempts on right and left sides. Mean of ordinal scores from 0: <= 10 cm to 10: >= 37 cm.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT. In the case of missing data, no replacement or imputation method was performed.
Measure: Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
centimeters
  Baseline | 20.18 [17.90 to 22.45] | 19.76 [17.64 to 21.87]
  Week 2 | 19.69 [17.36 to 22.03] | 18.81 [16.40 to 21.22]
  Week 4 | 19.19 [16.82 to 21.56] | 18.82 [16.54 to 21.09]
  Week 8 | 18.70 [16.39 to 21.01] | 20.03 [16.91 to 23.14]
  Week 12 | 18.54 [16.25 to 20.83] | 18.45 [16.06 to 20.83]

43. Secondary Outcome: Bath Ankylosing Spondylitis Metrology Index (BASMI): Spinal Mobility Measured With Tragus-to-wall Measurement at Weeks 14, 18, 24
Description: Measurement in centimeters (cm) of distance between the tragus and wall from right and left side while subject is standing with back against the wall; knees straight; scapulae, buttocks, and heels against the wall; with head in neutral position. Measurement of two tries on right and left sides. Mean of ordinal scores from 0: <= 10 cm to 10: >= 37 cm.
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; in the case of missing data, no replacement or imputation method was performed.
Measure: Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
centimeters
  Week 14 | 19.12 [16.86 to 21.38] | 18.38 [16.05 to 20.70]
  Week 18 | 19.86 [17.74 to 21.98] | 18.55 [16.17 to 20.94]
  Week 24 | 18.99 [16.85 to 21.13] | 18.60 [16.28 to 20.92]

44. Secondary Outcome: Bath Ankylosing Spondylitis Metrology Index (BASMI) Independent Component: Spinal Mobility Measured With Lateral Flexion at Baseline and Weeks 2, 4, 8, and 12
Description: Measurement in centimters (cm) of distance between subject's middle fingertip and the floor after bending sideways, without bending knees or lifting heels, while attemting to keep shoulders in same place (flexion position). Measurement of two attempts on each side (right and left). Mean of ordinal scores from 0: >=20 cm to 10: <=1.2 cm.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT. In the case of missing data, no replacement or imputation method was performed.
Measure: Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
centimeters
  Baseline | 13.79 [7.34 to 20.25] | 9.80 [5.30 to 14.30]
  Week 2 | 13.58 [7.57 to 19.59] | 10.62 [5.94 to 15.31]
  Week 4 | 13.01 [7.46 to 18.55] | 10.60 [5.75 to 15.45]
  Week 8 | 12.19 [6.74 to 17.63] | 10.21 [5.52 to 14.89]
  Week 12 | 12.41 [6.94 to 17.87] | 8.56 [4.41 to 12.71]

45. Secondary Outcome: Bath Ankylosing Spondylitis Metrology Index (BASMI): Spinal Mobility Measured With Lateral Flexion at Weeks 14, 18, 24
Description: Measurement in centimters (cm) of distance between subject's middle fingertip and the floor after bending sideways, without bending knees or lifting heels, while attempting to keep shoulders in same place (flexion position). Measurement of two attempts on each side (right and left). Mean of ordinal scores from 0: >=20 cm to 10: <=1.2 cm.
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; in the case of missing data, no replacement or imputation method was performed.
Measure: Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
centimeters
  Week 14 | 12.93 [7.41 to 18.44] | 8.19 [4.42 to 11.95]
  Week 18 | 12.02 [6.19 to 17.85] | 8.08 [4.85 to 11.31]
  Week 24 | 10.95 [6.47 to 15.44] | 10.48 [5.73 to 15.24]

46. Secondary Outcome: Bath Ankylosing Spondylitis Metrology Index (BASMI) Independent Component: Spinal Mobility Measured With Modified Schober's Test at Baseline and Weeks 2, 4, 8, 12
Description: Measurement in centimeters of the distance between marks originally placed while the subject was standing erect 10 centimeters (cm) above and 5 cm below the midpoint of a line that joints the posterior superior iliac spines. Distance between marks was remeasured with subject maximally bend forward, knees fully extended, with spine in full flexion. Measurement of two attempts. Mean of ordinal scores from 1: 5.7 to 6.3 cm, to 10: <=0.7 cm.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT. In the case of missing data, no replacement or imputation method was performed.
Measure: Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
centimeters
  Baseline | 1.63 [1.24 to 2.02] | 1.52 [1.10 to 1.93]
  Week 2 | 1.73 [1.28 to 2.18] | 1.57 [1.15 to 1.99]
  Week 4 | 1.85 [1.38 to 2.32] | 1.77 [1.28 to 2.26]
  Week 8 | 1.95 [1.47 to 2.42] | 1.57 [1.12 to 2.03]
  Week 12 | 1.88 [1.43 to 2.32] | 1.51 [1.05 to 1.97]

47. Secondary Outcome: Bath Ankylosing Spondylitis Metrology Index (BASMI): Spinal Mobility Measured With Modified Schober's Test at Weeks 14, 18, 24
Description: as for outcome 46
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; in the case of missing data, no replacement or imputation method was performed.
Measure: Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
centimeters
  Week 14 | 1.87 [1.39 to 2.36] | 1.63 [1.16 to 2.10]
  Week 18 | 1.71 [1.17 to 2.25] | 1.69 [1.21 to 2.17]
  Week 24 | 1.92 [1.41 to 2.44] | 1.79 [1.31 to 2.28]

48. Secondary Outcome: Bath Ankylosing Spondylitis Metrology Index (BASMI) Independent Component: Spinal Mobility Measured With Intermalleolar Distance at Baseline and Weeks 2, 4, 8, 12
Description: Measurement in centimeters (cm) of the distance between the medial malleoli when subject is lying supine with knees and feet straight up with legs separated as far as possible. Measurement of two attempts. Mean of ordinal scores from 0: >= 120 cm, to 9: 30 to 39.9 cm.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT. In the case of missing data, no replacement or imputation method was performed.
Measure: Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
centimeters
  Baseline | 82.31 [72.15 to 92.46] | 89.30 [81.60 to 97.00]
  Week 2 | 87.89 [78.83 to 96.94] | 92.08 [84.85 to 99.31]
  Week 4 | 90.86 [81.20 to 100.52] | 91.53 [82.97 to 100.08]
  Week 8 | 93.56 [85.19 to 101.92] | 91.58 [83.62 to 99.54]
  Week 12 | 94.46 [86.87 to 102.05] | 91.72 [83.84 to 99.60]

49. Secondary Outcome: Bath Ankylosing Spondylitis Metrology Index (BASMI): Spinal Mobility Measured With Intermalleolar Distance at Weeks 14, 18, 24
Description: as for outcome 48
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; in the case of missing data, no replacement or imputation method was performed.
Measure: Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
centimeters
  Week 14 | 95.79 [88.40 to 103.18] | 98.03 [90.25 to 105.81]
  Week 18 | 96.27 [88.76 to 103.78] | 96.66 [88.25 to 105.06]
  Week 24 | 95.71 [87.96 to 103.46] | 96.41 [88.86 to 103.95]

50. Secondary Outcome: Normalized Net Incremental Area Under the Curve (AUC) for the Chest Expansion Test Between Baseline and Week 12
Description: Normalized net incremental area under the curve (AUC) = area between baseline and the Chest Expansion Test curve as a function of time (randomization to Week 12); computed using the linear trapezoidal method. All areas above baseline and under the curve are positive and all areas below baseline and above the curve are negative. Net incremental AUC = sum of these areas; this result was then divided by the study duration of the patients; negative value = improvement.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF. N=number of subjects with evaluable data.
Measure: Least Squares Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 37 | 43
centimeters | 0.26 [0.05 to 0.48] | 0.19 [-0.01 to 0.39]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Analysis of covariance (ANCOVA) with treatment as a factor and baseline value as a covariate; Test type: Superiority or Other; p = 0.613, ANCOVA; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.22 to 0.37] — Least squares mean difference = mean difference final value

51. Secondary Outcome: Change From Baseline in the Chest Expansion Test at Weeks 2, 4, 8, 12
Description: Measurement and remeasurement of standing maximal inspiration; chest circumference at nipple line or at 4th intercostal space in centimeters.
Time Frame: Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF. N=number of subjects with evaluable data.
Measure: Least Squares Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 37 | 43
centimeters
  Week 2 | 0.17 [-0.12 to 0.46] | 0.10 [-0.17 to 0.38]
  Week 4 | 0.09 [-0.20 to 0.39] | 0.19 [-0.08 to 0.47]
  Week 8 | 0.43 [0.14 to 0.73] | 0.23 [-0.04 to 0.50]
  Week 12 | 0.39 [0.09 to 0.68] | 0.33 [0.05 to 0.60]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Week 2: mixed model analysis of covariance (ANCOVA), using an auto-regressive correlation structure, with treatment groups, visits, and their interaction as fixed factors, baseline value as a covariate and patients as a random factor; Test type: Superiority or Other; p = 0.744, ANCOVA; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.34 to 0.47] — Least squares mean difference = mean difference final value
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Week 4: mixed model analysis of covariance (ANCOVA), using an auto-regressive correlation structure, with treatment groups, visits, and their interaction as fixed factors, baseline value as a covariate and patients as a random factor; Test type: Superiority or Other; p = 0.625, ANCOVA; Mean Difference (Final Values) = -0.10, 95% CI [-0.50 to 0.30] — Least squares mean difference = mean difference final value
Statistical Analysis 3: Comparison: Etanercept vs Placebo; Week 8: mixed model analysis of covariance (ANCOVA), using an auto-regressive correlation structure, with treatment groups, visits, and their interaction as fixed factors, baseline value as a covariate and patients as a random factor; Test type: Superiority or Other; p = 0.325, ANCOVA; Mean Difference (Final Values) = 0.20, 95% CI [-0.20 to 0.60] — Least squares mean difference = mean difference final value
Statistical Analysis 4: Comparison: Etanercept vs Placebo; Week 12: mixed model analysis of covariance (ANCOVA), using an auto-regressive correlation structure, with treatment groups, visits, and their interaction as fixed factors, baseline value as a covariate and patients as a random factor; Test type: Superiority or Other; p = 0.760, ANCOVA; Mean Difference (Final Values) = 0.06, 95% CI [-0.34 to 0.46] — Least squares mean difference = mean difference final value

52. Secondary Outcome: Change From Baseline in the Chest Expansion Test at Weeks 14, 18, 24
Description: Measurement and remeasurement of standing maximal inspiration; chest circumference at nipple line or at 4th intercostal space in centimeters (cm).
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; LOCF.
Measure: Mean (95% Confidence Interval); unit: centimeters
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
centimeters
  Week 14 | 0.26 [-0.13 to 0.65] | 0.22 [-0.15 to 0.60]
  Week 18 | 0.22 [-0.16 to 0.60] | 0.33 [-0.08 to 0.75]
  Week 24 | 0.46 [0.01 to 0.90] | 0.44 [0.07 to 0.80]

53. Secondary Outcome: Change From Baseline in Level of Difficulty to Perform Physically Demanding Activities Due to Ankylosing Spondylitis at Weeks 2, 4, 8, 12
Description: Subject evaluation of level of difficulty to perform daily physical activities and/or kinesitherapy for ankylosing spondylitis (AS) because of AS using a 100 millimeter Visual Analog Scale (VAS) ranging from 0=easy to 100=impossible. Subgroup of subjects who responded that they were able to perform daily physical activities and/or kinesitherapy for their ankylosing spondylitis at each visit.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF. N = subgroup of subjects who reported performing daily physical activities and/or kinesitherapy for their ankylosing spondylitis at each visit (Week 2 through Week 12).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 18 | 17
units on scale
  Week 2 | -11.88 [-21.31 to -2.46] | -7.16 [-16.99 to 2.67]
  Week 4 | -15.14 [-24.67 to -5.60] | -12.04 [-21.77 to -2.32]
  Week 8 | -18.65 [-28.32 to -8.98] | -17.25 [-26.98 to -7.53]
  Week 12 | -22.55 [-32.19 to -12.91] | -18.53 [-28.37 to -8.69]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 38, analysis 1]; Test type: Superiority or Other; p = 0.490, ANCOVA; Mean Difference (Final Values) = -4.72, 95% CI 2-sided [-18.35 to 8.91] — Least squares mean difference = mean difference final value
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 38, analysis 2]; Test type: Superiority or Other; p = 0.651, ANCOVA; Mean Difference (Final Values) = -3.09, 95% CI [-16.73 to 10.54] — Least squares mean difference = mean difference final value
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 38, analysis 3]; Test type: Superiority or Other; p = 0.840, ANCOVA; Mean Difference (Final Values) = -1.39, 95% CI [-15.12 to 12.34] — Least squares mean difference = mean difference final value
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 38, analysis 4]; Test type: Superiority or Other; p = 0.562, ANCOVA; Mean Difference (Final Values) = -4.02, 95% CI [-17.81 to 9.77] — Least squares mean difference = mean difference final value

54. Secondary Outcome: Change From Baseline in Self Assessment of Ability and or Easiness to Perform Physically Demanding Activities at Weeks 14, 18, 24
Description: Subject evaluation of level of difficulty to perform daily physical activities and/or kinesitherapy for ankylosing spondylitis (AS) due to AS using a 100 millimeter Visual Analog Scale (VAS) ranging from 0=easy to 100=impossible. Subgroup of subjects who responded that they were able to perform daily physical activities and/or kinesitherapy for their ankylosing spondylitis at each visit.
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; LOCF.
Measure: Mean (95% Confidence Interval); unit: units on scale
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 17 | 17
units on scale
  Week 14 | -20.01 [-32.79 to -7.24] | -22.95 [-36.79 to -9.10]
  Week 18 | -22.39 [-35.92 to -8.86] | -27.80 [-42.80 to -12.81]
  Week 24 | -24.21 [-37.43 to -10.99] | -25.55 [-41.35 to -9.75]

55. Secondary Outcome: Normalized Net Incremental Area Under the Curve (AUC) for Erythtocyte Sedimentation Rate Between Baseline and Week 12
Description: Normalized net incremental area under the curve (AUC) = area between baseline and the Erythrocyte Sedimentation Rate curve as a function of time (randomization to Week 12); computed using the linear trapezoidal method. All areas above baseline and under the curve are positive and all areas below baseline and above the curve are negative. Net incremental AUC = sum of these areas; this result was then divided by the study duration of the patients; negative value = improvement.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF. N=number of subjects with evaluable data.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters per hour
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 42
millimeters per hour | -16.18 [-19.55 to -12.81] | -1.45 [-4.70 to 1.80]
Statistical Analysis 1: Comparison: Etanercept; Analysis of covariance (ANCOVA)with treatment as a factor and baseline vlue as a covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -14.73, 95% CI 2-sided [-19.44 to -10.03] — Least squares mean difference = mean difference final value

56. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Weeks 2, 4, 8, 12
Description: ESR is a laboratory test that provides a non-specific measure of inflammation. The test assesses the rate at which red blood cells fall in a test tube. A higher rate is consistent with inflammation.
Time Frame: Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF. N = number of subjects with evaluable data.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeters per hour
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 42
millimeters per hour
  Week 2 | -15.00 [-19.16 to -10.84] | -2.62 [-6.63 to 1.39]
  Week 4 | -20.05 [-24.21 to -15.89] | -2.60 [-6.61 to 1.41]
  Week 8 | -17.02 [-21.18 to -12.86] | -0.07 [-4.08 to 3.93]
  Week 12 | -20.33 [-24.49 to -16.17] | -2.17 [-6.18 to 1.84]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Week 2: Mixed model analysis of covariance (ANCOVA), using an auto-regressive correlation structure, with treatment groups, visits and their interaction as fixed factors, baseline value as a covariate and atients as a random factor; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -12.37, 95% CI 2-sided [-18.17 to -6.58] — Least squares mean difference = mean difference final value
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 38, analysis 2]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -17.45, 95% CI [-23.25 to -11.65] — Least squares mean difference = mean difference final value
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 38, analysis 3]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -16.95, 95% CI [-22.75 to -11.15] — Least squares mean difference = mean difference final value
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 38, analysis 4]; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -18.16, 95% CI [-23.96 to -12.36] — Least squares mean difference = mean difference final value

57. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Weeks 14, 18, 24
Description: as for outcome 56
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; LOCF.
Measure: Mean (95% Confidence Interval); unit: millimeters per hour
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
millimeters per hour
  Week 14 | -20.32 [-27.16 to -13.47] | -10.21 [-15.99 to -4.43]
  Week 18 | -17.95 [-25.50 to -10.39] | -12.32 [-17.45 to -7.18]
  Week 24 | -18.53 [-27.06 to -9.99] | -14.61 [-20.39 to -8.82]

58. Secondary Outcome: Normalized Net Incremental Area Under the Curve (AUC) for C-reactive Protein Between Baseline and Week 12
Description: Normalized net incremental area under the curve (AUC) = area between baseline and the C-reactive Protein curve as a function of time (randomization to Week 12); computed using the linear trapezoidal method. All areas above baseline and under the curve are positive and all areas below baseline and above the curve are negative. Net incremental AUC = sum of these areas; this result was then divided by the study duration of the patients; negative value = improvement.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT; LOCF.
Measure: Least Squares Mean (95% Confidence Interval); unit: milligrams per liter
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
milligrams per liter | -14.41 [-18.01 to -10.82] | -1.17 [-4.59 to 2.25]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Analysis of covariance (ANCOVA), with treatment as a factor and baseline value as a covariate; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -13.24, 95% CI 2-sided [-18.23 to -8.25] — Least squares mean difference = mean difference final value

59. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP) at Weeks 2, 4, 8, 12
Description: CRP is a marker of inflammation. A higher level is consistent with inflammation.
Time Frame: Baseline, Week 2, Week 4, Week 8, Week 12
Population: mITT. LOCF.
Measure: Least Squares Mean (95% Confidence Interval); unit: milligrams per liter
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
milligrams per liter
  Week 2 | -15.37 [-19.86 to -10.88] | -1.05 [-5.32 to 3.23]
  Week 4 | -16.99 [-21.48 to -12.50] | -2.01 [-6.28 to 2.26]
  Week 8 | -16.19 [-20.68 to -11.71] | -1.01 [-5.28 to 3.27]
  Week 12 | -15.69 [-20.18 to -11.20] | -1.28 [-5.55 to 2.99]
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Week 2: Mixed model analysis of covariance (ANCOVA), using an auto-regressive correlation structure, with treatment groups, visits and their interactions as fixed factors, baseline as a covariate and patients as a random factor; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -14.32, 95% CI 2-sided [-20.55 to -8.10] — Least squares mean difference = mean difference final value
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Week 4: Mixed model analysis of covariance (ANCOVA), using an auto-regressive correlation structure, with treatment groups, visits and their interactions as fixed factors, baseline as a covariate and patients as a random factor; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -14.98, 95% CI [-21.20 to -8.76] — Least squares mean difference = mean difference final value
Statistical Analysis 3: Comparison: Etanercept vs Placebo; Week 8: Mixed model analysis of covariance (ANCOVA), using an auto-regressive correlation structure, with treatment groups, visits and their interactions as fixed factors, baseline as a covariate and patients as a random factor; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -15.19, 95% CI [-21.41 to -8.96] — Least squares mean difference = mean difference final value
Statistical Analysis 4: Comparison: Etanercept vs Placebo; Week 12: Mixed model analysis of covariance (ANCOVA), using an auto-regressive correlation structure, with treatment groups, visits and their interactions as fixed factors, baseline as a covariate and patients as a random factor; Test type: Superiority or Other; p < 0.0001, ANCOVA; Mean Difference (Final Values) = -14.41, 95% CI [-20.63 to -8.19] — Least squares mean difference = mean difference final value

60. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP) at Weeks 14, 18, 24
Description: Change from baseline in C-reactive Protein (CRP).
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; LOCF.
Measure: Mean (95% Confidence Interval); unit: milligrams per liter
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
milligrams per liter
  Week 14 | -18.11 [-27.76 to -8.46] | -10.04 [-14.53 to -5.55]
  Week 18 | -17.15 [-26.73 to -7.58] | -9.47 [-13.19 to -5.75]
  Week 24 | -16.05 [-26.90 to -5.20] | -9.62 [-13.84 to -5.41]

61. Secondary Outcome: Percent of Subjects With Normal and Abnormal C-Reactive Protein at Weeks 14, 18, 24
Description: Percent of participants with normal (<6 milligrams per liter) and abnormal (>= 6 milligrams per liter) C-Reactive Protein.
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; LOCF.
Measure: Number; unit: percent of participants
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
percent of participants
  Week 14: Normal | 60.53 | 70.59
  Week 14: Abnormal | 39.47 | 29.41
  Week 18: Normal | 63.16 | 66.67
  Week 18: Abnormal | 36.84 | 33.33
  Week 24: Normal | 68.42 | 82.05
  Week 24: Abnormal | 31.58 | 17.95

62. Secondary Outcome: Percent of Subjects With Patient Acceptable and Unacceptable Symptom State (PASS) at Weeks 2, 4, 8, 12
Description: Percent of subjects reporting acceptable symptom state: acceptance to remain for the rest of their lives with the level of pain they had during the last 48 hours; and unacceptable symptom state: not able to remain for the rest of their lives with the level of pain they had during the last 48 hours. In the case of missing data, subjects who withdrew from the study because of inefficacy or toxicity were considered "unacceptable".
Time Frame: Week 2, Week 4, Week 8, Week 12
Population: mITT. In the case of missing data, no replacement or imputation method was performed.
Measure: Number; unit: percent of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
percent of participants
  Week 2: Acceptable | 43.24 | 30.00
  Week 2: Unacceptable | 56.76 | 70.00
  Week 4: Acceptable | 57.89 | 35.71
  Week 4: Unacceptable | 42.11 | 64.29
  Week 8: Acceptable | 68.42 | 33.33
  Week 8: Unacceptable | 31.58 | 66.67
  Week 12: Acceptable | 60.53 | 40.54
  Week 12: Unacceptable | 39.47 | 59.46
Statistical Analysis 1: Comparison: Etanercept vs Placebo; Week 2: Generalized estimating equation (GEE) model, using a logit link, binomial distribution and an auto-regressive correlation structure, with treatment groups, visits and their interaction as fixed factors; Test type: Superiority or Other; p = 0.184, GEE model; Odds Ratio (OR) = 1.87, 95% CI 2-sided [0.74 to 4.70] — An odds-ratio greater than 1 indicates the odds of response is greater in etanercept group than in placebo group
Statistical Analysis 2: Comparison: Etanercept vs Placebo; Week 4: Generalized estimating equation (GEE) model, using a logit link, binomial distribution and an auto-regressive correlation structure, with treatment groups, visits and their interaction as fixed factors; Test type: Superiority or Other; p = 0.036, GEE model; Odds Ratio (OR) = 2.62, 95% CI [1.06 to 6.46] — An odds-ratio greater than 1 indicates the odds of response is greater in etanercept group than in placebo group
Statistical Analysis 3: Comparison: Etanercept vs Placebo; Week 8: Generalized estimating equation (GEE) model, using a logit link, binomial distribution and an auto-regressive correlation structure, with treatment groups, visits and their interaction as fixed factors; Test type: Superiority or Other; p = 0.001, GEE model; Odds Ratio (OR) = 4.96, 95% CI [1.89 to 13.03] — An odds-ratio greater than 1 indicates the odds of response is greater in etanercept group than in placebo group
Statistical Analysis 4: Comparison: Etanercept vs Placebo; Week 12: Generalized estimating equation (GEE) model, using a logit link, binomial distribution and an auto-regressive correlation structure, with treatment groups, visits and their interaction as fixed factors; Test type: Superiority or Other; p = 0.065, GEE model; Odds Ratio (OR) = 2.38, 95% CI [0.95 to 5.96] — An odds-ratio greater than 1 indicates the odds of response is greater in etanercept group than in placebo group

63. Secondary Outcome: Percent of Subjects With Patient Acceptable and Unacceptable Symptom State (PASS) at Weeks 14, 18, 24
Description: as for outcome 62
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population. In the case of missing data, no replacement or imputation method was performed.
Measure: Number; unit: percent of participants
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
percent of participants
  Week 14: Acceptable | 69.44 | 64.71
  Week 14: Unacceptable | 30.56 | 35.29
  Week 18: Acceptable | 74.29 | 66.67
  Week 18: Unacceptable | 25.71 | 33.33
  Week 24: Acceptable | 77.14 | 80.56
  Week 24: Unacceptable | 22.86 | 19.44

64. Secondary Outcome: Percent of Subjects With Minimum Clinically Important Improvement (MCII) in Pain Rating at Weeks 2, 4, 8, 12
Description: Subjects were asked how their pain had been during the last 48 hours compared to baseline. Those subjects that reported improvement assessed how important this improvement was to them; range: very important, moderately important, slightly important, or not at all important. Binary response options: 1=improved very important, or improved moderately important; 2=slightly important, not at all important, no change, or worse-more pain.
Time Frame: Week 2, Week 4, Week 8, Week 12
Population: mITT; in the case of missing data, no replacement or imputation method was performed. Abbreviation: Mod = moderately.
Measure: Number; unit: percent of participants
Arm/Group | Etanercept | Placebo
Number analyzed (Participants) | 39 | 43
percent of participants
  Week 2: Improvement Very/Mod. Important | 50.00 | 20.00
  Week 2 : Improvement Slightly/Not Important | 50.00 | 80.00
  Week 4: Improvement Very/Mod. Important | 52.63 | 30.95
  Week 4: Improvement Slightly/Not Important | 47.37 | 69.05
  Week 8: Improvement Very/Mod. Important | 75.00 | 35.90
  Week 8: Improvement Slightly/Not Important | 25.00 | 64.10
  Week 12: Improvement Very/Mod. Important | 63.16 | 37.84
  Week 12: Improvement Slightly/Not Important | 36.84 | 62.16
Statistical Analysis 1: Comparison: Etanercept vs Placebo; [analysis description as in outcome 62, analysis 1]; Test type: Superiority or Other; p = 0.004, GEE model; Odds Ratio (OR) = 4.57, 95% CI 2-sided [1.64 to 12.74] — Odds ratio greater than 1 indicates the odds of response is greater in etanercept group than in placebo group
Statistical Analysis 2: Comparison: Etanercept vs Placebo; [analysis description as in outcome 62, analysis 2]; Test type: Superiority or Other; p = 0.054, GEE model; Odds Ratio (OR) = 2.46, 95% CI [0.99 to 6.12] — Odds ratio greater than 1 indicates the odds of response is greater in etanercept group than in placebo group
Statistical Analysis 3: Comparison: Etanercept vs Placebo; [analysis description as in outcome 62, analysis 3]; Test type: Superiority or Other; p < 0.001, GEE model; Odds Ratio (OR) = 6.26, 95% CI [2.27 to 17.31] — Odds ratio greater than 1 indicates the odds of response is greater in etanercept group than in placebo group
Statistical Analysis 4: Comparison: Etanercept vs Placebo; [analysis description as in outcome 62, analysis 4]; Test type: Superiority or Other; p = 0.025, GEE model; Odds Ratio (OR) = 2.88, 95% CI [1.14 to 7.27] — Odds ratio greater than 1 indicates the odds of response is greater in etanercept group than in placebo group

65. Secondary Outcome: Percent of Subjects With Minimum Clinially Important Improvement (MCII) at Weeks 14, 18, 24
Description: as for outcome 64
Time Frame: Week 14, Week 18, Week 24
Population: Open-label population; in the case of missing data, no replacement or imputation method was performed. Abbreviation: Mod = moderately.
Measure: Number; unit: percent of participants
Arm/Group | Etanercept/Etanercept | Placebo/Etanercept
Number analyzed (Participants) | 38 | 39
percent of participants
  Week 14: Improvement Very/Mod. Important | 77.78 | 77.14
  Week 14: Improvement Slightly/Not Important | 22.22 | 22.86
  Week 18: Improvement Very/Mod. Important | 94.12 | 78.38
  Week 18: Improvement Slightly/Not Important | 5.88 | 21.62
  Week 24: Improvement Very/Mod. Important | 91.43 | 86.11
  Week 24: Improvement Slightly/Not Important | 8.57 | 13.89

ADVERSE EVENTS:
Groups:
- Etanercept: Double-blind Period 1: Etanercept 50 mg subcutaneously (SC) once weekly
- Placebo: Double-blind Period 1: placebo subcutaneously (SC), once weekly
Arm/Group | Etanercept | Placebo | Etanercept/Etanercept | Placebo/Etanercept
Serious Adverse Events (participants affected / at risk) | 2/39 | 1/43 | 0/38 | 1/39
Other Adverse Events (participants affected / at risk) | 24/39 | 28/43 | 16/38 | 22/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=39) | Placebo (N=43) | Etanercept/Etanercept (N=38) | Placebo/Etanercept (N=39)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept (N=39) | Placebo (N=43) | Etanercept/Etanercept (N=38) | Placebo/Etanercept (N=39)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1
External ear pain (Ear and labyrinth disorders) | 1 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 0 | 0
Iridocyclitis (Eye disorders) | 1 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Asthenia (General disorders) | 1 | 1 | 0 | 0
Exercise tolerance decreased (General disorders) | 0 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 1
Injection site erythema (General disorders) | 2 | 0 | 0 | 0
Injection site haematoma (General disorders) | 1 | 0 | 0 | 0
Injection site pruritus (General disorders) | 1 | 0 | 1 | 2
Malaise (General disorders) | 0 | 1 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 1 | 0
Cytolytic hepatitis (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Seasonal allergy (Immune system disorders) | 0 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 2 | 1 | 1 | 1
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1 | 0 | 0
Hordeolum (Infections and infestations) | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 2 | 2
Otitis externa (Infections and infestations) | 0 | 1 | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 4 | 3 | 2 | 1
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 0
Tracheitis (Infections and infestations) | 1 | 0 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 3 | 2 | 2 | 1
Urinary tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0
Viral pharyngitis (Infections and infestations) | 0 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skeletal injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0
Haemoglobin urine present (Investigations) | 1 | 0 | 0 | 0
Transaminases increased (Investigations) | 3 | 1 | 0 | 0
Weight decreased (Investigations) | 0 | 1 | 0 | 0
Weight increased (Investigations) | 1 | 1 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Ankylosing spondylitis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 1 | 0
Headache (Nervous system disorders) | 2 | 3 | 0 | 0
Intercostal neuralgia (Nervous system disorders) | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0 | 0
Syncope vasovagal (Nervous system disorders) | 0 | 0 | 0 | 1
Trigeminal neuralgia (Nervous system disorders) | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Skin inflammation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 2
Hot flush (Vascular disorders) | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0 | 1
Lymphoedema (Vascular disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PIs agreed to allow the sponsor 60 days to review and require changes to presentations or publications but only to protect confidential information and intellectual property, and for the sponsor to file a patent application, as applicable. The PIs also agreed for data to be presented first as a joint, multi-center publication.